CLINICAL TRIAL: NCT04442737
Title: A Phase 4, Randomized, Active-Controlled, Open-label Study to Evaluate the Safety and Tolerability of Switching to Once-Daily Darunavir/Cobicistat/Emtricitabine/Tenofovir Alafenamide (D/C/F/TAF) Fixed-dose Combination (FDC) Regimen in Virologically-suppressed Human Immunodeficiency Virus Type 1 (HIV-1) Infected Participants Experiencing Rapid Weight Gain With an INI + TAF/FTC ARV Regimen
Brief Title: A Study of Darunavir/Cobicistat/Emtricitabine/Tenofovir Alafenamide (D/C/F/TAF) Evaluated as a Fixed Dose Combination Regimen in Participants Switching From an Integrase Inhibitor Who Have Experienced Rapid Weight Gain
Acronym: DEFINE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Janssen Scientific Affairs, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CR108757; TMC114FD2HTX4004 (Other: Janssen Scientific Affairs, LLC)
Record Dates: First submitted 2020-06-03; First posted 2020-06-23 (Actual); Results first posted 2024-08-27 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: HIV-1

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- D/C/F/TAF FDC Arm (Immediate Switch) (Experimental): Participants will be immediately switched to a regimen of darunavir 800 milligram (mg)/cobicistat 150 mg/emtricitabine 200 mg/tenofovir alafenamide 10 mg (D/C/F/TAF) fixed-dose combination (FDC) once daily for 48 weeks.
  Interventions: Drug: D/C/F/TAF FDC
- INI + TAF/FTC Arm (Delayed Switch) (Active Comparator): Participants will continue to receive current baseline integrase (INI)-based regimen plus Tenofovir Alafenamide/Emtricitabine (TAF/FTC) antiretroviral (ARV) regimen for 24 weeks. After 24 weeks participants will switch to a regimen of D/C/F/TAF FDC once daily for an additional 24 weeks.
  Interventions: Drug: D/C/F/TAF FDC; Drug: TAF/FTC FDC; Drug: INI Based Regimen

INTERVENTIONS:
Drug: D/C/F/TAF FDC — A FDC tablet containing darunavir 800 mg, cobicistat 150 mg, emtricitabine 200 mg, tenofovir alafenamide 10 mg will be administered once daily.
Drug: TAF/FTC FDC — TAF/FTC ARV regimen will be administered once daily.
  Arms: INI + TAF/FTC Arm (Delayed Switch)
Drug: INI Based Regimen — The integrase (INI) inhibitors (for example, bictegravir, dolutegravir, elvitegravir/cobicistat, and raltegravir) will be administered in combination with TAF/FTC, as appropriate. Regimen may consist of a single tablet regimen or a combination of two separate pills.
  Arms: INI + TAF/FTC Arm (Delayed Switch)

SUMMARY:
The purpose of this study is to assess the percent change in body weight when switching to darunavir/cobicistat/emtricitabine/tenofovir alafenamide (D/C/F/TAF) fixed-dose combination (FDC) (Immediate Switch Arm) compared to continuing the current integrase (INI) + tenofovir alafenamide/emtricitabine (TAF/FTC) antiretroviral (ARV) regimen (Delayed Switch Arm) in virologically-suppressed human immunodeficiency virus (HIV)-1 infected participants who have experienced rapid and significant body weight gain.

ELIGIBILITY:
Inclusion Criteria:

* Body Mass Index (BMI) of greater than or equal to (>=) 18 kilogram per meter square (kg/m^2) at time of starting an integrase (INI)-based regimen plus Tenofovir Alafenamide/Emtricitabine (TAF/FTC) antiretroviral (ARV) regimen
* Documented human immunodeficiency virus (HIV)-1 infection
* Currently being treated with a stable ARV regimen consisting of an INI combined with TAF/FTC for >=6 consecutive months preceding the screening visit and experienced a >=10 percent (%) increase in body weight within a 36-month time period prior to screening and while on the current INI + TAF/FTC ARV regimen
* Documented evidence of being virologically suppressed while on the current stable INI+TAF/FTC ARV regimen prior to screening
* At least one plasma HIV-1 RNA measurement less than (<) 50 copies/milliliter (mL) occurring between 12 and 2 months prior to the screening visit while on the stable INI+ TAF/FTC ARV regimen and have HIV-1 RNA <50 copies/ mL at the screening visit

Exclusion Criteria:

* Known history of malignancy within the past 5 years or ongoing malignancy other than cutaneous Kaposi's sarcoma, basal cell carcinoma, or resected, noninvasive cutaneous squamous carcinoma
* Known allergies, hypersensitivity, or intolerance to D/C/F/TAF fixed-dose combination (FDC) tablet or its excipients
* Active hepatitis B (HBV) or hepatitis C virus (HCV) infection
* Uncontrolled diabetes that will require treatment with insulin during the study period
* Evidence of Child Pugh Class C based on clinical laboratory testing and clinical evaluation
* History of failure on darunavir (DRV) treatment or known documented history of >=1 DRV resistance-associated mutations (RAM)
* Screening hepatic transaminases >5x the upper limit of the normal range
* Screening creatinine based estimated glomerular filtration rate (eGFRcr) <30 ml/min according to the Cockcroft-Gault formula for creatinine clearance
* Participants initiating or discontinuing concomitant medications associated with significant changes in weight within the last 90 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 103 (Actual)
Dates: Start 2020-07-01 (Actual); Primary Completion 2023-08-07 (Actual); Study Completion 2023-08-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Scientific Affairs, LLC Clinical Trial, Study Director — Janssen Scientific Affairs, LLC
Locations (34):
- United States (34):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - The Office of Franco Felizarta, MD, Bakersfield, California
  - AIDS Health Foundation-Westside HCC, Beverly Hills, California
  - Long Beach Education & Research Consultants, Long Beach, California
  - Midway Immunology and Research Center, Ft. Pierce, Florida
  - University of Miami, Miami, Florida
  - Triple O Research Institute, West Palm Beach, Florida
  - Atlanta ID Group, Atlanta, Georgia
  - Medical College of Georgia, Augusta, Georgia
  - The Corporation of Mercer University, Macon, Georgia
  - Chatham County Health Department, Savannah, Georgia
  - The Ruth M. Rothstein CORE Center, Chicago, Illinois
  - Care South Clinic, Baton Rouge, Louisiana
  - Kaiser Permanente, Rockville, Maryland
  - Community Research Initiative, Boston, Massachusetts
  - Be Well Medical Center, PC, Berkley, Michigan
  - Henry Ford Health System, Detroit, Michigan
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Washington University School Of Medicine, St Louis, Missouri
  - University of Nebraska, Omaha, Nebraska
  - Saint Michaels Medical Center - Infectious Disease, Newark, New Jersey
  - AIDS Healthcare Foundation-Research Center, New York, New York
  - Mount Sinai Hospital-New York, New York, New York
  - Montefiore Medical Center, The Bronx, New York
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Philadelphia Fight, Philadelphia, Pennsylvania
  - Palmetto Health - USC, Columbia, South Carolina
  - AIDS Arms Incorporated Trinity Health and Wellness Center, Dallas, Texas
  - North Texas Infectious Diseases Consultants, Dallas, Texas
  - Texas Centers for Infectious Disease Associates, Fort Worth, Texas
  - Therapeutic Concepts - Donald R Watkins Foundation, Houston, Texas
  - DCOL Center for Clinical Research, Longview, Texas
  - Infectious Disease Associates of Central Virginia, Lynchburg, Virginia
  - Vivent Health, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of the Janssen Pharmaceutical Companies of Johnson & Johnson is available at www.janssen.com/clinical-trials/transparency. As noted on this site, requests for access to the study data can be submitted through Yale open Data Access (YODA) Project site at yoda.yale.edu
URL: https://www.janssen.com/clinical-trials/transparency

REFERENCES:
- [Derived] Anderson D, Ramgopal M, Hagins DP, Lee J, Simonson RB, Hsu TH, Xu P, Ahmad N, Short WR. DEFINE: A Prospective, Randomized, Phase 4 Trial to Assess a Protease Inhibitor-Based Regimen Switch Strategy to Manage Integrase Inhibitor-Related Weight Gain. Clin Infect Dis. 2025 Mar 17;80(3):602-612. doi: 10.1093/cid/ciae449. PMID 39230668

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: As per change in planned analysis, data for resistance outcome measures were not collected and analyzed due to insufficient number of participants who met the criteria for virologic rebound/failure.
Groups:
- D/C/F/TAF Immediate Switch (IS): Baseline to Week 48: Virologically suppressed adult participants with >=10% increase in weight within 36 month period prior to screening and while on current integrase (INI) inhibitor along with tenofovir alafenamide 10 mg, emtricitabine 200 mg (TAF/FTC) antiretroviral (ARV) (INI + TAF/FTC ARV) regimen switched to receive a fixed-dose combination (FDC) regimen of darunavir 800 milligrams (mg), cobicistat 150 mg, emtricitabine 200 mg, and tenofovir alafenamide 10 mg (D/C/F/TAF), once daily from Day 1 (baseline) up to Week 48.
- INI + TAF/FTC Delayed Switch (DS): Baseline to Week 48: Virologically suppressed adult participants with >=10% increase in weight within 36 month period prior to screening and while on current INI + TAF/FTC ARV regimen continued to receive baseline integrase (INI) inhibitor along with tenofovir alafenamide 10 mg, emtricitabine 200 mg (TAF/FTC) antiretroviral (ARV) regimen from baseline up to Week 24 per prescribing information (delayed switch 1 [DS1]). After Week 24, participants switched to receive D/C/F/TAF FDC once daily from Week 25 to Week 48 (DS2).
Period: Overall Study
Arm/Group | D/C/F/TAF Immediate Switch (IS): Baseline to Week 48 | INI + TAF/FTC Delayed Switch (DS): Baseline to Week 48
Started | 53 | 50
Treatment Phase IS1: Baseline up to Week 24 | 53 | 0
Treatment Phase IS2: Week 25 to Week 48 | 49 | 0
Treatment Phase DS1: Baseline up to Week 24 | 0 | 50
Treatment Phase DS2: Week 25 to Week 48 | 0 | 49
Completed | 45 | 39
Not Completed | 8 | 11
Not completed — Lost to Follow-up | 1 | 3
Not completed — Withdrawal by Subject | 3 | 2
Not completed — Adverse Event | 3 | 2
Not completed — Death | 0 | 1
Not completed — Protocol Violation | 0 | 2
Not completed — Other | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | D/C/F/TAF Immediate Switch (IS): Baseline to Week 48 | INI + TAF/FTC Delayed Switch (DS): Baseline to Week 48 | Total
Number analyzed (Participants) | 53 | 50 | 103
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.5 (12.27) | 46.1 (11.7) | 43.7 (12.16)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 15 | 31
  Male | 37 | 35 | 72
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 10 | 16
  Not Hispanic or Latino | 47 | 40 | 87
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 33 | 30 | 63
  White | 19 | 19 | 38
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 1 | 0 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States of America | 53 | 50 | 103

OUTCOME MEASURES:

1. Primary Outcome: Percent Change From Baseline in Body Weight at Week 24
Description: Percent change from baseline in body weight at Week 24 were reported.
Time Frame: Baseline and Week 24
Population: The intent-to-treat (ITT) analysis set included all the participants who were randomized and received at least 1 dose of treatment subsequent to randomization in the study. Here, 'N' (number of participants analyzed) signifies number of participants evaluable for this outcome measure.
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent Change
Groups:
- D/C/F/TAF Immediate Switch (IS1): Baseline to Week 24: Virologically suppressed adult participants with >=10% increase in weight within 36 month period prior to screening and while on current INI + TAF/FTC ARV regimen switched to receive a fixed-dose combination (FDC) regimen of darunavir 800 milligrams (mg), cobicistat 150 mg, emtricitabine 200 mg, and tenofovir alafenamide 10 mg (D/C/F/TAF), once daily from Day 1 (baseline) up to Week 24.
- INI + TAF/FTC Delayed Switch (DS1): Baseline to Week 24: Virologically suppressed adult participants with >=10% increase in weight within 36 month period prior to screening and while on current INI + TAF/FTC ARV regimen continued to receive baseline integrase (INI) inhibitor along with tenofovir alafenamide 10 mg, emtricitabine 200 mg (TAF/FTC) antiretroviral (ARV) regimen from Day 1 (baseline) up to Week 24 per prescribing information (delayed switch 1 [DS1]).
Arm/Group | D/C/F/TAF Immediate Switch (IS1): Baseline to Week 24 | INI + TAF/FTC Delayed Switch (DS1): Baseline to Week 24
Number analyzed (Participants) | 49 | 46
Percent Change | 0.63 [-0.435 to 1.698] | -0.24 [-1.354 to 0.874]

2. Primary Outcome: Percent Change From Baseline in Body Weight at Week 24: Body Mass Index (BMI) >=30 Kilograms Per Square Meter (kg/m^2) Subgroup
Description: Percent change from baseline in body weight at Week 24 in BMI >=30 kilograms per square meter (kg/m^2) subgroup were reported.
Time Frame: Baseline and Week 24
Population: The ITT analysis set included all the participants who were randomized and received at least 1 dose of treatment subsequent to randomization in the study. Here, 'N' (number of participants analyzed) signifies number of participants evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: Percent Change
Arm/Group | D/C/F/TAF Immediate Switch (IS1): Baseline to Week 24 | INI + TAF/FTC Delayed Switch (DS1): Baseline to Week 24
Number analyzed (Participants) | 26 | 36
Percent Change | 0.26 (4.278) | 0.18 (3.247)

3. Primary Outcome: Percent Change From Baseline in Body Weight at Week 24: Female and Male Subgroup
Description: Percent change from baseline in body weight at Week 24 in female and male subgroup were reported.
Time Frame: Baseline and Week 24
Population: The ITT analysis set included all the participants who were randomized and received at least 1 dose of treatment subsequent to randomization in the study. Here, 'N' (number of participants analyzed) signifies number of participants evaluable for this outcome measure. Here, 'n' (number analyzed) is defined as participants analyzed at specified categories.
Measure: Mean (Standard Deviation); unit: Percent Change
Arm/Group | D/C/F/TAF Immediate Switch (IS1): Baseline to Week 24 | INI + TAF/FTC Delayed Switch (DS1): Baseline to Week 24
Number analyzed (Participants) | 49 | 46
Percent Change
  Female Subgroup: number analyzed (Participants) | 14 | 15
  Female Subgroup | 1.26 (5.361) | -0.89 (2.632)
  Male Subgroup: number analyzed (Participants) | 35 | 31
  Male Subgroup | 0.46 (3.939) | -0.22 (6.609)

4. Primary Outcome: Percent Change From Baseline in Body Weight at Week 24: Black/African American and Black/African American- Female Subgroups
Description: Percent change from baseline in body weight at Week 24 in Black/African American and Black/African American- Female subgroups were reported.
Time Frame: Baseline and Week 24
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Percent Change
Arm/Group | D/C/F/TAF Immediate Switch (IS1): Baseline to Week 24 | INI + TAF/FTC Delayed Switch (DS1): Baseline to Week 24
Number analyzed (Participants) | 30 | 29
Percent Change
  Black/African American Subgroups | 0.50 (5.043) | -1.36 (5.925)
  Black/African American- Female Subgroups: number analyzed (Participants) | 12 | 12
  Black/African American- Female Subgroups | 0.62 (5.484) | -0.82 (2.894)

5. Primary Outcome: Percent Change From Baseline in Body Weight at Week 24: Non-Black/African American Subgroup
Description: Percent change from baseline in body weight at Week 24 in Non-Black/African American subgroup were reported.
Time Frame: Baseline and Week 24
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Percent Change
Arm/Group | D/C/F/TAF Immediate Switch (IS1): Baseline to Week 24 | INI + TAF/FTC Delayed Switch (DS1): Baseline to Week 24
Number analyzed (Participants) | 19 | 17
Percent Change | 1.00 (3.045) | 1.14 (4.756)

6. Secondary Outcome: Change From Baseline in Absolute Body Weight Over Time
Description: Change from baseline in absolute body weight over time were reported.
Time Frame: INI + TAF/FTC Delayed Switch (DS1) and D/C/F/TAF Immediate Switch (IS1): Baseline, Weeks 4, 12, 24; D/C/F/TAF Immediate Switch (IS): Baseline, Week 36 and 48
Population: The ITT analysis set included all the participants who were randomized and received at least 1 dose of treatment subsequent to randomization in the study. Here, 'N' (number of participants analyzed) is number of participants evaluable for this outcome measure. Here, 'n' (number analyzed) is defined as participants analyzed at specified timepoints. Here, n=0 signifies that participants were not planned to be analyzed at those timepoints in the respective arms.
Measure: Median (Inter-Quartile Range); unit: Kilograms (kg)
Groups:
- D/C/F/TAF Immediate Switch (IS1): Baseline to Week 24: Virologically suppressed adult participants with >=10% increase in weight within 36 month period prior to screening and while on current integrase (INI) inhibitor along with tenofovir alafenamide 10 mg, emtricitabine 200 mg (TAF/FTC) antiretroviral (ARV) (INI + TAF/FTC ARV) regimen switched to receive a fixed-dose combination (FDC) regimen of darunavir 800 milligrams (mg), cobicistat 150 mg, emtricitabine 200 mg, and tenofovir alafenamide 10 mg (D/C/F/TAF), once daily from Day 1 (baseline) up to Week 24.
Arm/Group | INI + TAF/FTC Delayed Switch (DS1): Baseline to Week 24 | D/C/F/TAF Immediate Switch (IS1): Baseline to Week 24 | D/C/F/TAF Immediate Switch (IS): Baseline to Week 48
Number analyzed (Participants) | 49 | 53 | 47
Kilograms (kg)
  Week 4: number analyzed (Participants) | 49 | 53 | 0
  Week 4 | -0.20 [-1.10 to 0.70] | -0.20 [-1.50 to 0.90] |
  Week 12: number analyzed (Participants) | 45 | 52 | 0
  Week 12 | 0.10 [-1.20 to 2.30] | 0.20 [-2.35 to 1.55] |
  Week 24: number analyzed (Participants) | 46 | 49 | 0
  Week 24 | 0.30 [-2.10 to 2.30] | 0.50 [-2.30 to 2.60] |
  Week 36: number analyzed (Participants) | 0 | 0 | 47
  Week 36 |  |  | -0.90 [-3.40 to 2.10]
  Week 48: number analyzed (Participants) | 0 | 0 | 46
  Week 48 |  |  | -0.85 [-4.50 to 1.70]

7. Secondary Outcome: Percentage of Participants With Change From Baseline Greater Than or Equal to (>=) 3% to <= 5% in Body Weight Over Time
Description: Percentage of participants with change from baseline >=3% to <= 5% in body weight over time was reported.
Time Frame: as for outcome 6
Population: The ITT analysis set included all the participants who were randomized and received at least 1 dose of treatment subsequent to randomization in the study. Here, n=0 signifies that participants were not planned to be analyzed at those timepoints in the respective arms.
Measure: Number; unit: Percentage of Participants
Arm/Group | INI + TAF/FTC Delayed Switch (DS1): Baseline to Week 24 | D/C/F/TAF Immediate Switch (IS1): Baseline to Week 24 | D/C/F/TAF Immediate Switch (IS): Baseline to Week 48
Number analyzed (Participants) | 50 | 53 | 53
Percentage of Participants
  3-5% gain: Week 4: number analyzed (Participants) | 50 | 53 | 0
  3-5% gain: Week 4 | 2.0 | 3.8 |
  3-5% loss: Week 4: number analyzed (Participants) | 50 | 53 | 0
  3-5% loss: Week 4 | 4.1 | 7.5 |
  3-5% gain: Week 12: number analyzed (Participants) | 50 | 53 | 0
  3-5% gain: Week 12 | 8.9 | 5.8 |
  3-5% loss: Week 12: number analyzed (Participants) | 50 | 53 | 0
  3-5% loss: Week 12 | 4.4 | 17.3 |
  3-5% gain: Week 24: number analyzed (Participants) | 50 | 53 | 0
  3-5% gain: Week 24 | 2.2 | 8.2 |
  3-5% loss: Week 24: number analyzed (Participants) | 50 | 53 | 0
  3-5% loss: Week 24 | 8.7 | 10.2 |
  3-5% gain: Week 36: number analyzed (Participants) | 0 | 0 | 53
  3-5% gain: Week 36 |  |  | 6.4
  3-5% loss: Week 36: number analyzed (Participants) | 0 | 0 | 53
  3-5% loss: Week 36 |  |  | 14.9
  3-5% gain: Week 48: number analyzed (Participants) | 0 | 0 | 53
  3-5% gain: Week 48 |  |  | 6.5
  3-5% loss: Week 48: number analyzed (Participants) | 0 | 0 | 53
  3-5% loss: Week 48 |  |  | 6.5

8. Secondary Outcome: Percentage of Participants With Change From Baseline Greater Than (>) 5 Percent (%) in Body Weight Over Time
Description: Percentage of participants with change from baseline >5% in body weight over time was reported.
Time Frame: as for outcome 6
Population: as for outcome 7
Measure: Number; unit: Percentage of Participants
Arm/Group | INI + TAF/FTC Delayed Switch (DS1): Baseline to Week 24 | D/C/F/TAF Immediate Switch (IS1): Baseline to Week 24 | D/C/F/TAF Immediate Switch (IS): Baseline to Week 48
Number analyzed (Participants) | 50 | 53 | 53
Percentage of Participants
  >5% gain: Week 4: number analyzed (Participants) | 50 | 53 | 0
  >5% gain: Week 4 | 4.1 | 0 |
  >5% loss: Week 4: number analyzed (Participants) | 50 | 53 | 0
  >5% loss: Week 4 | 2.0 | 0 |
  >5% gain: Week 12: number analyzed (Participants) | 50 | 53 | 0
  >5% gain: Week 12 | 6.7 | 3.8 |
  >5% loss: Week 12: number analyzed (Participants) | 50 | 53 | 0
  >5% loss: Week 12 | 4.4 | 1.9 |
  >5% gain: Week 24: number analyzed (Participants) | 50 | 53 | 0
  >5% gain: Week 24 | 10.9 | 14.3 |
  >5% loss: Week 24: number analyzed (Participants) | 50 | 53 | 0
  >5% loss: Week 24 | 10.9 | 4.1 |
  >5% gain: Week 36: number analyzed (Participants) | 0 | 0 | 53
  >5% gain: Week 36 |  |  | 17.0
  >5% loss: Week 36: number analyzed (Participants) | 0 | 0 | 53
  >5% loss: Week 36 |  |  | 14.9
  >5% gain: Week 48: number analyzed (Participants) | 0 | 0 | 53
  >5% gain: Week 48 |  |  | 13.0
  >5% loss: Week 48: number analyzed (Participants) | 0 | 0 | 53
  >5% loss: Week 48 |  |  | 23.9

9. Secondary Outcome: Change From Baseline in Body Mass Index (BMI) Over Time
Description: Change from baseline in BMI over time was reported. BMI was calculated as weight (kg)/(height (m^2).
Time Frame: as for outcome 6
Population: as for outcome 6
Measure: Median (Inter-Quartile Range); unit: Kilograms per meter square (kg/m^2)
Arm/Group | INI + TAF/FTC Delayed Switch (DS1): Baseline to Week 24 | D/C/F/TAF Immediate Switch (IS1): Baseline to Week 24 | D/C/F/TAF Immediate Switch (IS): Baseline to Week 48
Number analyzed (Participants) | 49 | 53 | 47
Kilograms per meter square (kg/m^2)
  Week 4: number analyzed (Participants) | 49 | 53 | 0
  Week 4 | -0.06 [-0.35 to 0.22] | -0.07 [-0.51 to 0.27] |
  Week 12: number analyzed (Participants) | 45 | 52 | 0
  Week 12 | 0.03 [-0.42 to 0.75] | 0.07 [-0.78 to 0.50] |
  Week 24: number analyzed (Participants) | 46 | 49 | 0
  Week 24 | 0.10 [-0.66 to 0.77] | 0.20 [-0.67 to 0.80] |
  Week 36: number analyzed (Participants) | 0 | 0 | 47
  Week 36 |  |  | -0.26 [-1.17 to 0.70]
  Week 48: number analyzed (Participants) | 0 | 0 | 46
  Week 48 |  |  | -0.26 [-1.42 to 0.66]

10. Secondary Outcome: Change From Baseline in Body Composition as Measured by Dual-energy X-ray Absorptiometry (DEXA) Scan at Weeks 24 and 48
Description: Change from baseline in body composition as measured by (DEXA) scan at Weeks 24 and 48 was reported. Body composition included Mass of Fat for Trunk, Lean Body Mass for Trunk, total Mass for Trunk, Mass of Fat for Total Body, Lean Body Mass for Total Body, Total Mass for Total Body, Mass of Fat for Adjusted Total Body, Lean Body Mass for Adjusted Total Body, Total Mass for Adjusted Total Body, Mass of Fat for Appendages, Lean Body Mass for Appendages, total Mass for Appendages, Mass of Visceral Adipose Tissue, and Volume of Visceral Adipose Tissue. Adjusted refers to not including participant's head.
Time Frame: INI + TAF/FTC Delayed Switch (DS1): Baseline, Week 24; D/C/F/TAF Immediate Switch (IS1): Baseline, Week 24; D/C/F/TAF Immediate Switch (IS): Baseline, Week 48
Population: as for outcome 6
Measure: Median (Inter-Quartile Range); unit: Kilograms (kg)
Arm/Group | INI + TAF/FTC Delayed Switch (DS1): Baseline to Week 24 | D/C/F/TAF Immediate Switch (IS1): Baseline to Week 24 | D/C/F/TAF Immediate Switch (IS): Baseline to Week 48
Number analyzed (Participants) | 29 | 29 | 27
Kilograms (kg)
  Mass of Fat for Trunk: Week 24: number analyzed (Participants) | 29 | 29 | 0
  Mass of Fat for Trunk: Week 24 | -0.59 [-1.50 to 0.41] | 0.12 [-0.96 to 1.14] |
  Mass of Fat for Trunk: Week 48: number analyzed (Participants) | 0 | 0 | 27
  Mass of Fat for Trunk: Week 48 |  |  | -1.24 [-2.03 to 0.54]
  Lean Body Mass for Trunk: Week 24: number analyzed (Participants) | 29 | 29 | 0
  Lean Body Mass for Trunk: Week 24 | -0.51 [-1.19 to 0.45] | 0.22 [-0.89 to 0.83] |
  Lean Body Mass for Trunk: Week 48: number analyzed (Participants) | 0 | 0 | 27
  Lean Body Mass for Trunk: Week 48 |  |  | -0.29 [-1.08 to 1.11]
  Total Mass for Trunk: Week 24: number analyzed (Participants) | 29 | 29 | 0
  Total Mass for Trunk: Week 24 | -0.84 [-2.12 to 0.80] | 0.26 [-0.90 to 1.09] |
  Total Mass for Trunk: Week 48: number analyzed (Participants) | 0 | 0 | 27
  Total Mass for Trunk: Week 48 |  |  | -1.41 [-1.99 to 0.57]
  Mass of Fat for Total Body: Week 24: number analyzed (Participants) | 29 | 29 | 0
  Mass of Fat for Total Body: Week 24 | -0.88 [-2.75 to 0.62] | 0.29 [-1.45 to 1.77] |
  Mass of Fat for Total Body: Week 48: number analyzed (Participants) | 0 | 0 | 27
  Mass of Fat for Total Body: Week 48 |  |  | -1.29 [-3.20 to 1.18]
  Lean Body Mass for Total Body: Week 24: number analyzed (Participants) | 29 | 29 | 0
  Lean Body Mass for Total Body: Week 24 | 0.22 [-2.44 to 1.50] | 0.52 [-1.27 to 1.76] |
  Lean Body Mass for Total Body: Week 48: number analyzed (Participants) | 0 | 0 | 27
  Lean Body Mass for Total Body: Week 48 |  |  | -0.42 [-2.18 to 1.16]
  Total Mass for Total Body: Week 24: number analyzed (Participants) | 29 | 29 | 0
  Total Mass for Total Body: Week 24 | 0.22 [-3.21 to 2.57] | 0.59 [-0.61 to 2.04] |
  Total Mass for Total Body: Week 48: number analyzed (Participants) | 0 | 0 | 27
  Total Mass for Total Body: Week 48 |  |  | -1.32 [-3.93 to 0.24]
  Mass of Fat for Adjusted Total Body: Week 24: number analyzed (Participants) | 29 | 29 | 0
  Mass of Fat for Adjusted Total Body: Week 24 | -0.88 [-2.71 to 0.68] | 0.41 [-1.44 to 1.76] |
  Mass of Fat for Adjusted Total Body: Week 48: number analyzed (Participants) | 0 | 0 | 27
  Mass of Fat for Adjusted Total Body: Week 48 |  |  | -1.28 [-3.16 to 1.26]
  Lean Body Mass for Adjusted Total Body: Week 24: number analyzed (Participants) | 29 | 29 | 0
  Lean Body Mass for Adjusted Total Body: Week 24 | 0.17 [-2.34 to 1.58] | 0.49 [-1.30 to 2.01] |
  Lean Body Mass for Adjusted Total Body: Week 48: number analyzed (Participants) | 0 | 0 | 27
  Lean Body Mass for Adjusted Total Body: Week 48 |  |  | -0.38 [-2.25 to 1.17]
  Total Mass for Adjusted Total Body: Week 24: number analyzed (Participants) | 29 | 29 | 0
  Total Mass for Adjusted Total Body: Week 24 | -0.01 [-3.23 to 2.42] | 0.56 [-0.66 to 2.03] |
  Total Mass for Adjusted Total Body: Week 48: number analyzed (Participants) | 0 | 0 | 27
  Total Mass for Adjusted Total Body: Week 48 |  |  | -1.43 [-3.98 to 0.14]
  Mass of Fat for Appendages: Week 24: number analyzed (Participants) | 29 | 29 | 0
  Mass of Fat for Appendages: Week 24 | 0.00 [-1.30 to 0.45] | 0.34 [-0.14 to 0.69] |
  Mass of Fat for Appendages: Week 48: number analyzed (Participants) | 0 | 0 | 27
  Mass of Fat for Appendages: Week 48 |  |  | -0.52 [-1.41 to 0.40]
  Lean Body Mass for Appendages: Week 24: number analyzed (Participants) | 29 | 29 | 0
  Lean Body Mass for Appendages: Week 24 | 0.72 [-0.65 to 1.30] | 0.12 [-1.06 to 0.89] |
  Lean Body Mass for Appendages: Week 48: number analyzed (Participants) | 0 | 0 | 27
  Lean Body Mass for Appendages: Week 48 |  |  | -0.32 [-0.81 to 0.27]
  Total Mass for Appendages: Week 24: number analyzed (Participants) | 29 | 29 | 0
  Total Mass for Appendages: Week 24 | 0.66 [-1.38 to 1.90] | 0.46 [-0.59 to 1.55] |
  Total Mass for Appendages: Week 48: number analyzed (Participants) | 0 | 0 | 27
  Total Mass for Appendages: Week 48 |  |  | -0.69 [-1.70 to 0.31]
  Mass of Visceral Adipose Tissue: Week 24: number analyzed (Participants) | 26 | 29 | 0
  Mass of Visceral Adipose Tissue: Week 24 | -0.05 [-0.14 to 0.12] | 0.03 [-0.06 to 0.14] |
  Mass of Visceral Adipose Tissue: Week 48: number analyzed (Participants) | 0 | 0 | 27
  Mass of Visceral Adipose Tissue: Week 48 |  |  | -0.05 [-0.11 to 0.04]

11. Secondary Outcome: Change From Baseline in Waist Circumference Over Time
Description: Change from baseline in waist circumference over time was reported.
Time Frame: as for outcome 6
Population: as for outcome 6
Measure: Median (Inter-Quartile Range); unit: Centimeter (cm)
Arm/Group | INI + TAF/FTC Delayed Switch (DS1): Baseline to Week 24 | D/C/F/TAF Immediate Switch (IS1): Baseline to Week 24 | D/C/F/TAF Immediate Switch (IS): Baseline to Week 48
Number analyzed (Participants) | 49 | 53 | 47
Centimeter (cm)
  Week 4: number analyzed (Participants) | 49 | 53 | 0
  Week 4 | 0.00 [-3.00 to 0.80] | 0.00 [-2.50 to 1.50] |
  Week 12: number analyzed (Participants) | 45 | 52 | 0
  Week 12 | 0.20 [-1.00 to 2.50] | 0.00 [-2.00 to 2.70] |
  Week 24: number analyzed (Participants) | 46 | 49 | 0
  Week 24 | 0.00 [-5.10 to 2.50] | 0.80 [-3.30 to 4.00] |
  Week 36: number analyzed (Participants) | 0 | 0 | 47
  Week 36 |  |  | 0.00 [-2.00 to 3.80]
  Week 48: number analyzed (Participants) | 0 | 0 | 46
  Week 48 |  |  | -0.40 [-4.90 to 4.10]

12. Secondary Outcome: Change From Baseline in Systolic Blood Pressure (SBP) and Diastolic Blood Pressure (DBP) Over Time
Description: Change from baseline in SBP and DBP over time was reported.
Time Frame: as for outcome 6
Population: as for outcome 6
Measure: Median (Inter-Quartile Range); unit: Milligrams of mercury (mmHg)
Arm/Group | INI + TAF/FTC Delayed Switch (DS1): Baseline to Week 24 | D/C/F/TAF Immediate Switch (IS1): Baseline to Week 24 | D/C/F/TAF Immediate Switch (IS): Baseline to Week 48
Number analyzed (Participants) | 49 | 53 | 47
Milligrams of mercury (mmHg)
  SBP: Week 4: number analyzed (Participants) | 49 | 53 | 0
  SBP: Week 4 | 3.0 [-7.0 to 9.0] | -2.0 [-10.0 to 7.0] |
  SBP: Week 12: number analyzed (Participants) | 45 | 52 | 0
  SBP: Week 12 | 0.0 [-5.0 to 6.0] | 1.0 [-9.0 to 6.0] |
  SBP: Week 24: number analyzed (Participants) | 46 | 49 | 0
  SBP: Week 24 | 0.5 [-8.0 to 7.0] | -3.0 [-9.0 to 5.0] |
  SBP: Week 36: number analyzed (Participants) | 0 | 0 | 47
  SBP: Week 36 |  |  | -5.0 [-11.0 to 5.0]
  SBP: Week 48: number analyzed (Participants) | 0 | 0 | 46
  SBP: Week 48 |  |  | -3.0 [-11.0 to 10.0]
  DBP: Week 4: number analyzed (Participants) | 49 | 47 | 0
  DBP: Week 4 | 0.0 [-3.0 to 4.0] | -2.0 [-8.0 to 3.0] |
  DBP: Week 12: number analyzed (Participants) | 45 | 52 | 0
  DBP: Week 12 | -1.0 [-5.0 to 4.0] | -2.0 [-7.0 to 3.5] |
  DBP: Week 24: number analyzed (Participants) | 46 | 49 | 0
  DBP: Week 24 | 0.0 [-4.0 to 4.0] | 0.0 [-6.0 to 4.0] |
  DBP: Week 36: number analyzed (Participants) | 0 | 0 | 47
  DBP: Week 36 |  |  | -2.0 [-9.0 to 3.0]
  DBP: Week 48: number analyzed (Participants) | 0 | 0 | 46
  DBP: Week 48 |  |  | -2.5 [-8.0 to 2.0]

13. Secondary Outcome: Change From Baseline in Fasting Lipids at Weeks 24 and 48
Description: Change from baseline in fasting lipids at Weeks 24 and 48 was reported. Fasting lipids included: fasting total cholesterol, fasting high-density lipoprotein (HDLs) and low-density lipoprotein (LDLs), and fasting triglycerides.
Time Frame: as for outcome 10
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: millimoles per liter (mmol/L)
Arm/Group | INI + TAF/FTC Delayed Switch (DS1): Baseline to Week 24 | D/C/F/TAF Immediate Switch (IS1): Baseline to Week 24 | D/C/F/TAF Immediate Switch (IS): Baseline to Week 48
Number analyzed (Participants) | 41 | 43 | 44
millimoles per liter (mmol/L)
  Fasting total cholesterol: Week 24: number analyzed (Participants) | 41 | 43 | 0
  Fasting total cholesterol: Week 24 | 0.11 (0.847) | 0.86 (0.790) |
  Fasting total cholesterol: Week 48: number analyzed (Participants) | 0 | 0 | 44
  Fasting total cholesterol: Week 48 |  |  | 0.73 (0.828)
  Fasting HDL: Week 24: number analyzed (Participants) | 41 | 42 | 0
  Fasting HDL: Week 24 | -0.13 (0.337) | 0.04 (0.269) |
  Fasting HDL: Week 48: number analyzed (Participants) | 0 | 0 | 44
  Fasting HDL: Week 48 |  |  | 0.05 (0.321)
  Fasting LDL: Week 24: number analyzed (Participants) | 41 | 42 | 0
  Fasting LDL: Week 24 | 0.15 (0.758) | 0.57 (0.768) |
  Fasting LDL: Week 48: number analyzed (Participants) | 0 | 0 | 44
  Fasting LDL: Week 48 |  |  | 0.59 (0.791)
  Fasting triglycerides: Week 24: number analyzed (Participants) | 41 | 42 | 0
  Fasting triglycerides: Week 24 | 0.16 (0.575) | 0.49 (0.902) |
  Fasting triglycerides: Week 48: number analyzed (Participants) | 0 | 0 | 44
  Fasting triglycerides: Week 48 |  |  | 0.28 (0.832)

14. Secondary Outcome: Change From Baseline in Fasting Glucose at Weeks 24 and 48
Description: Change from baseline in fasting glucose at Weeks 24 and 48 was reported.
Time Frame: as for outcome 10
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | INI + TAF/FTC Delayed Switch (DS1): Baseline to Week 24 | D/C/F/TAF Immediate Switch (IS1): Baseline to Week 24 | D/C/F/TAF Immediate Switch (IS): Baseline to Week 48
Number analyzed (Participants) | 42 | 43 | 45
mmol/L
  Week 24: number analyzed (Participants) | 42 | 43 | 0
  Week 24 | 0.05 (0.933) | -0.08 (0.697) |
  Week 48: number analyzed (Participants) | 0 | 0 | 45
  Week 48 |  |  | 0.06 (0.663)

15. Secondary Outcome: Change From Baseline in Homeostatic Model Assessment of Insulin Resistance (HOMA-IR) at Weeks 24 and 48
Description: Change from baseline in HOMA-IR at Weeks 24 and 48 was reported. HOMA-IR is calculated as fasting insulin * fasting glucose divided by 405.
Time Frame: as for outcome 10
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: Milligrams per deciliter (mg/dL)
Arm/Group | INI + TAF/FTC Delayed Switch (DS1): Baseline to Week 24 | D/C/F/TAF Immediate Switch (IS1): Baseline to Week 24 | D/C/F/TAF Immediate Switch (IS): Baseline to Week 48
Number analyzed (Participants) | 43 | 47 | 44
Milligrams per deciliter (mg/dL)
  Week 24: number analyzed (Participants) | 43 | 47 | 0
  Week 24 | -0.81 (7.946) | -0.05 (6.699) |
  Week 48: number analyzed (Participants) | 0 | 0 | 44
  Week 48 |  |  | 0.01 (7.164)

16. Secondary Outcome: Change From Baseline in Percent of Hemoglobin A1c (HbA1c) at Weeks 24 and 48
Description: Change from baseline in percent of HbA1c at Weeks 24 and 48 was reported.
Time Frame: as for outcome 10
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: Percent of HbA1c
Arm/Group | INI + TAF/FTC Delayed Switch (DS1): Baseline to Week 24 | D/C/F/TAF Immediate Switch (IS1): Baseline to Week 24 | D/C/F/TAF Immediate Switch (IS): Baseline to Week 48
Number analyzed (Participants) | 44 | 46 | 46
Percent of HbA1c
  Week 24: number analyzed (Participants) | 44 | 46 | 0
  Week 24 | 0.01 (0.272) | -0.07 (0.308) |
  Week 48: number analyzed (Participants) | 0 | 0 | 46
  Week 48 |  |  | -0.10 (0.313)

17. Secondary Outcome: Change From Baseline in Leptin at Weeks 24 and 48
Description: Change from baseline in leptin at Weeks 24 and 48 was reported.
Time Frame: as for outcome 10
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: Micrograms per liter (mcg/L)
Arm/Group | INI + TAF/FTC Delayed Switch (DS1): Baseline to Week 24 | D/C/F/TAF Immediate Switch (IS1): Baseline to Week 24 | D/C/F/TAF Immediate Switch (IS): Baseline to Week 48
Number analyzed (Participants) | 41 | 35 | 39
Micrograms per liter (mcg/L)
  Week 24: number analyzed (Participants) | 41 | 35 | 0
  Week 24 | -6.85 (16.077) | -1.09 (10.899) |
  Week 48: number analyzed (Participants) | 0 | 0 | 39
  Week 48 |  |  | 4.11 (22.787)

18. Secondary Outcome: Change From Baseline in Adiponectin at Weeks 24 and 48
Description: Change from baseline in adiponectin at Weeks 24 and 48 was reported.
Time Frame: as for outcome 10
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: Micrograms per liter (mcg/L)
Arm/Group | INI + TAF/FTC Delayed Switch (DS1): Baseline to Week 24 | D/C/F/TAF Immediate Switch (IS1): Baseline to Week 24 | D/C/F/TAF Immediate Switch (IS): Baseline to Week 48
Number analyzed (Participants) | 45 | 44 | 44
Micrograms per liter (mcg/L)
  Week 24: number analyzed (Participants) | 45 | 44 | 0
  Week 24 | -0.16 (1.596) | -0.11 (1.229) |
  Week 48: number analyzed (Participants) | 0 | 0 | 44
  Week 48 |  |  | 0.05 (1.589)

19. Secondary Outcome: Percentage of Participants With Advanced Fibrosis as Assessed by Non-alcoholic Fatty Liver Disease (NAFLD) Fibrosis Score at Weeks 24 and 48
Description: Percentage of participants with advanced fibrosis as assessed by NAFLD fibrosis score at Week 24 and 48 was reported. The NAFLD is based on a combination of clinical and laboratory measurements (that is, age, glycemia, BMI, platelet, albumin and AST/ALT ratio). The set cutoffs for this scoring are: NAFLD Score <-1.455 = F0-F2 (negative), NAFLD Score -1.455 to 0.675 = indeterminate score, NAFLD Score >0.675 = F3 - F4 (positive). NAFLD score was calculated as: 1.675 + 0.037 * age (years) + 0.094 * BMI (kg/m^2) + 1.13 * Impaired Fasting Glucose or Diabetes (yes =1; no=0) + 0.99 * AST/ALT ratio minus 0.013 * platelet (10^9/L) minus 0.66 * albumin (g/dL).
Time Frame: INI + TAF/FTC Delayed Switch (DS1) and D/C/F/TAF Immediate Switch (IS1): Week 24; D/C/F/TAF Immediate Switch (IS): Week 48
Population: The ITT analysis set included all the participants who were randomized and received at least 1 dose of treatment subsequent to randomization in the study. Here, 'N' (number of participants analyzed) is number of participants evaluable for this outcome measure. Here, n=0 signifies that participants were not planned to be analyzed at those timepoints in the respective arms.
Measure: Number; unit: Percentage of Participants
Arm/Group | INI + TAF/FTC Delayed Switch (DS1): Baseline to Week 24 | D/C/F/TAF Immediate Switch (IS1): Baseline to Week 24 | D/C/F/TAF Immediate Switch (IS): Baseline to Week 48
Number analyzed (Participants) | 50 | 53 | 53
Percentage of Participants
  Negative (F0-F2): Week 24: number analyzed (Participants) | 50 | 53 | 0
  Negative (F0-F2): Week 24 | 44.0 | 50.9 |
  Negative (F0-F2): Week 48: number analyzed (Participants) | 0 | 0 | 53
  Negative (F0-F2): Week 48 |  |  | 54.7
  Indeterminate: Week 24: number analyzed (Participants) | 50 | 53 | 0
  Indeterminate: Week 24 | 5.7 | 12.0 |
  Indeterminate: Week 48: number analyzed (Participants) | 0 | 0 | 53
  Indeterminate: Week 48 |  |  | 9.4
  Positive (F3-F4): Week 24: number analyzed (Participants) | 50 | 53 | 0
  Positive (F3-F4): Week 24 | 6.0 | 5.7 |
  Positive (F3-F4): Week 48: number analyzed (Participants) | 0 | 0 | 53
  Positive (F3-F4): Week 48 |  |  | 1.9

20. Secondary Outcome: Percentage of Participants at High Risk of Non-alcoholic Fatty Liver Disease (NASH) According to the Hypertension, Age, Insulin, Resistance (HAIR) Score at Weeks 24 and 48
Description: Percentage of participants at high risk of NASH according to the HAIR score at Weeks 24 and 48 was reported. HAIR score (0-3) is calculated by adding Hypertension = 1, alanine aminotransferase (ALT) >40 international unit (IU)=1, and Insulin resistance index (IR) >5.0 = 1. A score of >=2 is considered as high risk for NASH.
Time Frame: as for outcome 10
Population: as for outcome 19
Measure: Number; unit: Percentage of Participants
Arm/Group | INI + TAF/FTC Delayed Switch (DS1): Baseline to Week 24 | D/C/F/TAF Immediate Switch (IS1): Baseline to Week 24 | D/C/F/TAF Immediate Switch (IS): Baseline to Week 48
Number analyzed (Participants) | 50 | 53 | 53
Percentage of Participants
  <2: Week 24: number analyzed (Participants) | 50 | 53 | 0
  <2: Week 24 | 62.0 | 60.4 |
  <2: Week 48: number analyzed (Participants) | 0 | 0 | 53
  <2: Week 48 |  |  | 56.6
  >=2: Week 24: number analyzed (Participants) | 50 | 53 | 0
  >=2: Week 24 | 12.0 | 3.8 |
  >=2: Week 48: number analyzed (Participants) | 0 | 0 | 53
  >=2: Week 48 |  |  | 5.7

21. Secondary Outcome: Percentage of Participants With a Dose-reduction or Complete Withdrawal of Anti-hypertensive, Anti-hyperglycemic, or Lipid Lowering Agents
Description: Percentage of participants with a dose-reduction or complete withdrawal of anti-hypertensive, anti-hyperglycemic, or lipid lowering agents were reported.
Time Frame: D/C/F/TAF Immediate Switch (IS1) and INI + TAF/FTC Delayed Switch (DS1): Baseline up to Week 24; D/C/F/TAF Immediate Switch (IS2) and INI + TAF/FTC to D/C/F/TAF Delayed Switch (DS2): Week 25 up to Week 48
Population: The safety analysis set included all randomized participants who received at least 1 dose of study intervention (that is, ITT analysis set).
Measure: Number; unit: Percentage of Participants
Groups:
- D/C/F/TAF Immediate Switch (IS1): Baseline-Week 24: Virologically suppressed adult participants with >=10% increase in weight within 36 month period prior to screening and while on current INI + TAF/FTC ARV regimen switched to receive a fixed-dose combination (FDC) regimen of darunavir 800 milligrams (mg), cobicistat 150 mg, emtricitabine 200 mg, and tenofovir alafenamide 10 mg (D/C/F/TAF), once daily from Day 1 (baseline) up to Week 24.
- D/C/F/TAF Immediate Switch (IS2): Week 25-48: Virologically suppressed adult participants with >=10% increase in weight within 36 month period prior to screening and while on current INI + TAF/FTC ARV regimen switched to receive a fixed-dose combination (FDC) regimen of darunavir 800 milligrams (mg), cobicistat 150 mg, emtricitabine 200 mg, and tenofovir alafenamide 10 mg (D/C/F/TAF), once daily from Day 25 up to Week 48.
- INI + TAF/FTC to D/C/F/TAF Delayed Switch (DS2): Week 25-Week 48: Virologically suppressed adult participants with >=10% increase in weight within 36 month period prior to screening and while on current INI + TAF/FTC ARV regimen, after Week 24 switched to receive D/C/F/TAF FDC once daily from Week 25 to Week 48 (DS2).
Arm/Group | D/C/F/TAF Immediate Switch (IS1): Baseline-Week 24 | D/C/F/TAF Immediate Switch (IS2): Week 25-48 | INI + TAF/FTC Delayed Switch (DS1): Baseline to Week 24 | INI + TAF/FTC to D/C/F/TAF Delayed Switch (DS2): Week 25-Week 48
Number analyzed (Participants) | 53 | 49 | 50 | 46
Percentage of Participants
  Anti-hypertensive | 0 | 0 | 0 | 0
  Anti-hyperglycemic agents | 0 | 0. | 0 | 0
  Lipid lowering agents | 0 | 0 | 0 | 0

22. Secondary Outcome: Percentage of Participants Initiating an Anti-hypertensive, Anti-hyperglycemic, or Lipid Lowering Agents
Description: Percentage of participants initiating an anti-hypertensive, anti-hyperglycemic, or lipid lowering agents were reported.
Time Frame: as for outcome 21
Population: as for outcome 21
Measure: Number; unit: Percentage of Participants
Arm/Group | D/C/F/TAF Immediate Switch (IS1): Baseline-Week 24 | D/C/F/TAF Immediate Switch (IS2): Week 25-48 | INI + TAF/FTC Delayed Switch (DS1): Baseline to Week 24 | INI + TAF/FTC to D/C/F/TAF Delayed Switch (DS2): Week 25-Week 48
Number analyzed (Participants) | 53 | 49 | 50 | 46
Percentage of Participants
  Anti-hypertensive | 7.5 | 5.7 | 18.0 | 12.0
  Anti-hyperglycemic agents | 0 | 0. | 4.0 | 2.0
  Lipid lowering agents | 3.8 | 1.9 | 4.0 | 4.0

23. Secondary Outcome: Number of Participants With Any Grade Treatment-emergent Adverse Events (TEAEs)
Description: Number of participants with any grade TEAEs was reported. An AE is any untoward medical event that occurs in a participants administered an investigational product, and it does not necessarily indicate only events with clear causal relationship with the relevant investigational product. TEAEs were those AE events that occurred at or after the initial administration of study intervention.
Time Frame: as for outcome 21
Population: as for outcome 21
Measure: Count of Participants; unit: Participants
Arm/Group | D/C/F/TAF Immediate Switch (IS1): Baseline-Week 24 | INI + TAF/FTC Delayed Switch (DS1): Baseline to Week 24 | D/C/F/TAF Immediate Switch (IS2): Week 25-48 | INI + TAF/FTC to D/C/F/TAF Delayed Switch (DS2): Week 25-Week 48
Number analyzed (Participants) | 53 | 50 | 49 | 46
Participants | 30 | 29 | 26 | 30

24. Secondary Outcome: Number of Participants With Grade 3 and Grade 4 TEAEs
Description: Number of participants with Grade 3 and Grade 4 TEAEs were reported. An AE is any untoward medical event that occurs in a participants administered an investigational product, and it does not necessarily indicate only events with clear causal relationship with the relevant investigational product. TEAEs were those AE events that occurred at or after the initial administration of study intervention. Grades were assessed by Division of Acquired Immunodeficiency Syndrome (DAIDS) grading table: Grade 1: mild event; Grade 2: moderate event; Grade 3: severe event; Grade 4: potentially life-threatening event; Grade 5: death. Higher grades indicated worsening of TEAEs.
Time Frame: as for outcome 21
Population: as for outcome 21
Measure: Count of Participants; unit: Participants
Arm/Group | INI + TAF/FTC Delayed Switch (DS1): Baseline to Week 24 | D/C/F/TAF Immediate Switch (IS1): Baseline-Week 24 | D/C/F/TAF Immediate Switch (IS2): Week 25-48 | INI + TAF/FTC to D/C/F/TAF Delayed Switch (DS2): Week 25-Week 48
Number analyzed (Participants) | 50 | 53 | 49 | 46
Participants
  Grade 3 | 3 | 3 | 3 | 5
  Grade 4 | 0 | 1 | 0 | 1

25. Secondary Outcome: Number of Participants Who Discontinued the Study Drug Due to TEAEs
Description: Number of participants who discontinued the study drug due to TEAEs were reported. An AE is any untoward medical event that occurs in a participants administered an investigational product, and it does not necessarily indicate only events with clear causal relationship with the relevant investigational product. TEAEs were those AE events that occurred at or after the initial administration of study intervention.
Time Frame: as for outcome 21
Population: as for outcome 21
Measure: Count of Participants; unit: Participants
Arm/Group | INI + TAF/FTC Delayed Switch (DS1): Baseline to Week 24 | D/C/F/TAF Immediate Switch (IS1): Baseline-Week 24 | D/C/F/TAF Immediate Switch (IS2): Week 25-48 | INI + TAF/FTC to D/C/F/TAF Delayed Switch (DS2): Week 25-Week 48
Number analyzed (Participants) | 50 | 53 | 49 | 46
Participants | 0 | 3 | 0 | 2

26. Secondary Outcome: Number of Participants With Treatment-emergent Serious Adverse Events (SAEs)
Description: Number of participants with treatment-emergent SAEs were reported. An AE is any untoward medical occurrence in a participant participating in a clinical study that does not necessarily have a causal relationship with the pharmaceutical/biological agent under study. An SAE is an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly/birth defect; suspected transmission of any infectious agent via a medicinal product or medically important. Treatment-emergent SAEs were those SAE events that occurred at or after the initial administration of study intervention.
Time Frame: as for outcome 21
Population: as for outcome 21
Measure: Count of Participants; unit: Participants
Arm/Group | INI + TAF/FTC Delayed Switch (DS1): Baseline to Week 24 | D/C/F/TAF Immediate Switch (IS1): Baseline-Week 24 | D/C/F/TAF Immediate Switch (IS2): Week 25-48 | INI + TAF/FTC to D/C/F/TAF Delayed Switch (DS2): Week 25-Week 48
Number analyzed (Participants) | 50 | 53 | 49 | 46
Participants | 4 | 3 | 2 | 4

27. Secondary Outcome: Change From Baseline in Biochemistry Parameters: Albumin and Protein Values at Weeks 24 and 48
Description: Change from baseline in biochemistry parameters: albumin and protein values at Weeks 24 and 48 were reported.
Time Frame: as for outcome 10
Population: The safety analysis set included all randomized participants who received at least 1 dose of study intervention (that is, ITT analysis set). Here, 'N' (number of participants analyzed) is number of participants evaluable for this outcome measure. Here, 'n' (number analyzed) is defined as participants analyzed at specified timepoints. Here, n=0 signifies that participants were not planned to be analyzed at those timepoints in the respective arms.
Measure: Mean (Standard Deviation); unit: grams per liter (g/L)
Arm/Group | INI + TAF/FTC Delayed Switch (DS1): Baseline to Week 24 | D/C/F/TAF Immediate Switch (IS1): Baseline to Week 24 | D/C/F/TAF Immediate Switch (IS): Baseline to Week 48
Number analyzed (Participants) | 43 | 46 | 46
grams per liter (g/L)
  Albumin: Week 24: number analyzed (Participants) | 43 | 44 | 0
  Albumin: Week 24 | 0.1 (3.21) | 0.4 (2.17) |
  Albumin: Week 48: number analyzed (Participants) | 0 | 0 | 46
  Albumin: Week 48 |  |  | 0.1 (2.43)
  Protein: Week 24: number analyzed (Participants) | 43 | 44 | 0
  Protein: Week 24 | -0.4 (3.88) | 1.8 (3.53) |
  Protein: Week 48: number analyzed (Participants) | 0 | 0 | 46
  Protein: Week 48 |  |  | 0.6 (3.64)

28. Secondary Outcome: Change From Baseline in Biochemistry Parameters: Alkaline Phosphatase, Alanine Aminotransferase, and Aspartate Aminotransferase Values at Weeks 24 and 48
Description: Change from baseline in biochemistry parameters: Alkaline Phosphatase, Alanine Aminotransferase, and Aspartate Aminotransferase values at Weeks 24 and 48 were reported.
Time Frame: as for outcome 10
Population: as for outcome 27
Measure: Mean (Standard Deviation); unit: units per liter (U/L)
Arm/Group | INI + TAF/FTC Delayed Switch (DS1): Baseline to Week 24 | D/C/F/TAF Immediate Switch (IS1): Baseline to Week 24 | D/C/F/TAF Immediate Switch (IS): Baseline to Week 48
Number analyzed (Participants) | 43 | 44 | 46
units per liter (U/L)
  Alkaline Phosphatase: Week 24: number analyzed (Participants) | 43 | 44 | 0
  Alkaline Phosphatase: Week 24 | 8.50 (1.30) | 0.0 (10.84) |
  Alkaline Phosphatase: Week 48: number analyzed (Participants) | 0 | 0 | 46
  Alkaline Phosphatase: Week 48 |  |  | -2.8 (14.33)
  Alanine Aminotransferase: Week 24: number analyzed (Participants) | 43 | 44 | 0
  Alanine Aminotransferase: Week 24 | -4.2 (17.15) | -3.7 (10.96) |
  Alanine Aminotransferase: Week 48: number analyzed (Participants) | 0 | 0 | 46
  Alanine Aminotransferase: Week 48 |  |  | -0.1 (29.60)
  Aspartate Aminotransferase: Week 24: number analyzed (Participants) | 42 | 44 | 0
  Aspartate Aminotransferase: Week 24 | -4.2 (19.35) | -2.6 (6.66) |
  Aspartate Aminotransferase: Week 48: number analyzed (Participants) | 0 | 0 | 45
  Aspartate Aminotransferase: Week 48 |  |  | -1.6 (11.77)

29. Secondary Outcome: Change From Baseline in Biochemistry Parameters: Bicarbonate, Calcium, Cholesterol, Chloride, Potassium, Phosphate, Sodium, Triglycerides, and Urea Nitrogen Values at Weeks 24 and 48
Description: Change from baseline in biochemistry parameters: Bicarbonate, Calcium, Cholesterol, Chloride, Potassium, Phosphate, Sodium, Triglycerides, and Urea Nitrogen values at Weeks 24 and 48 were reported.
Time Frame: as for outcome 10
Population: as for outcome 27
Measure: Mean (Standard Deviation); unit: millimoles per liter (mmol/L)
Arm/Group | INI + TAF/FTC Delayed Switch (DS1): Baseline to Week 24 | D/C/F/TAF Immediate Switch (IS1): Baseline to Week 24 | D/C/F/TAF Immediate Switch (IS): Baseline to Week 48
Number analyzed (Participants) | 43 | 46 | 46
millimoles per liter (mmol/L)
  Bicarbonate: Week 24: number analyzed (Participants) | 43 | 43 | 0
  Bicarbonate: Week 24 | 0.70 (2.624) | 0.09 (2.661) |
  Bicarbonate: Week 48: number analyzed (Participants) | 0 | 0 | 43
  Bicarbonate: Week 48 |  |  | 0.52 (2.685)
  Calcium: Week 24: number analyzed (Participants) | 43 | 44 | 0
  Calcium: Week 24 | 0.00 (0.097) | 0.02 (0.092) |
  Calcium: Week 48: number analyzed (Participants) | 0 | 0 | 46
  Calcium: Week 48 |  |  | -0.02 (0.099)
  Cholesterol: Week 24: number analyzed (Participants) | 42 | 44 | 0
  Cholesterol: Week 24 | 0.11 (0.839) | 0.86 (0.782) |
  Cholesterol: Week 48: number analyzed (Participants) | 0 | 0 | 45
  Cholesterol: Week 48 |  |  | 0.72 (0.823)
  Chloride: Week 24: number analyzed (Participants) | 43 | 46 | 0
  Chloride: Week 24 | -0.4 (3.13) | -1.1 (3.07) |
  Chloride: Week 48: number analyzed (Participants) | 0 | 0 | 46
  Chloride: Week 48 |  |  | -0.8 (3.05)
  Potassium: Week 24: number analyzed (Participants) | 43 | 44 | 0
  Potassium: Week 24 | -0.07 (0.296) | -0.03 (0.421) |
  Potassium: Week 48: number analyzed (Participants) | 0 | 0 | 46
  Potassium: Week 48 |  |  | -0.10 (0.425)
  Phosphate: Week 24: number analyzed (Participants) | 43 | 44 | 0
  Phosphate: Week 24 | 0.01 (0.199) | -0.06 (0.166) |
  Phosphate: Week 48: number analyzed (Participants) | 0 | 0 | 46
  Phosphate: Week 48 |  |  | -0.05 (0.213)
  Sodium: Week 24: number analyzed (Participants) | 43 | 44 | 0
  Sodium: Week 24 | 0.1 (3.47) | -1.0 (2.89) |
  Sodium: Week 48: number analyzed (Participants) | 0 | 0 | 46
  Sodium: Week 48 |  |  | -0.7 (2.68)
  Triglycerides: Week 24: number analyzed (Participants) | 42 | 43 | 0
  Triglycerides: Week 24 | 0.13 (0.593) | 0.47 (0.898) |
  Triglycerides: Week 48: number analyzed (Participants) | 0 | 0 | 45
  Triglycerides: Week 48 |  |  | 0.26 (0.826)
  Urea Nitrogen: Week 24: number analyzed (Participants) | 43 | 44 | 0
  Urea Nitrogen: Week 24 | -0.05 (1.187) | 0.04 (1.240) |
  Urea Nitrogen: Week 48: number analyzed (Participants) | 0 | 0 | 46
  Urea Nitrogen: Week 48 |  |  | -0.27 (1.245)

30. Secondary Outcome: Change From Baseline in Hematology Parameters: Basophils, Eosinophils, Lymphocytes, Monocytes, Neutrophils (Segmented), Platelets, and Leukocytes Values at Weeks 24 and 48
Description: Change from baseline in hematology parameters: Basophils, Eosinophils, Lymphocytes, Monocytes, Neutrophils (segmented), Platelets, and Leukocytes values at Weeks 24 and 48 were reported.
Time Frame: as for outcome 10
Population: as for outcome 27
Measure: Mean (Standard Deviation); unit: 10^9 cells per liter
Arm/Group | INI + TAF/FTC Delayed Switch (DS1): Baseline to Week 24 | D/C/F/TAF Immediate Switch (IS1): Baseline to Week 24 | D/C/F/TAF Immediate Switch (IS): Baseline to Week 48
Number analyzed (Participants) | 43 | 45 | 45
10^9 cells per liter
  Basophils: Week 24: number analyzed (Participants) | 43 | 42 | 0
  Basophils: Week 24 | 0.00 (0.032) | 0.00 (0.036) |
  Basophils: Week 48: number analyzed (Participants) | 0 | 0 | 45
  Basophils: Week 48 |  |  | -0.01 (0.024)
  Eosinophils: Week 24: number analyzed (Participants) | 43 | 42 | 0
  Eosinophils: Week 24 | -0.01 (0.070) | -0.01 (0.104) |
  Eosinophils: Week 48: number analyzed (Participants) | 0 | 0 | 45
  Eosinophils: Week 48 |  |  | -0.02 (0.063)
  Lymphocytes: Week 24: number analyzed (Participants) | 43 | 42 | 0
  Lymphocytes: Week 24 | 0.04 (0.631) | -0.15 (0.517) |
  Lymphocytes: Week 48: number analyzed (Participants) | 0 | 0 | 45
  Lymphocytes: Week 48 |  |  | -0.17 (0.459)
  Monocytes: Week 24: number analyzed (Participants) | 43 | 42 | 0
  Monocytes: Week 24 | -0.02 (0.117) | 0.00 (0.094) |
  Monocytes: Week 48: number analyzed (Participants) | 0 | 0 | 45
  Monocytes: Week 48 |  |  | -0.01 (0.105)
  Neutrophils (segmented): Week 24: number analyzed (Participants) | 43 | 42 | 0
  Neutrophils (segmented): Week 24 | 0.04 (1.254) | 0.11 (1.144) |
  Neutrophils (segmented): Week 48: number analyzed (Participants) | 0 | 0 | 45
  Neutrophils (segmented): Week 48 |  |  | -0.04 (0.759)
  Platelets: Week 24: number analyzed (Participants) | 43 | 45 | 0
  Platelets: Week 24 | 2.0 (30.65) | -9.1 (38.58) |
  Platelets: Week 48: number analyzed (Participants) | 0 | 0 | 45
  Platelets: Week 48 |  |  | -8.5 (41.67)
  Leukocytes: Week 24: number analyzed (Participants) | 43 | 42 | 0
  Leukocytes: Week 24 | 0.05 (1.599) | -0.06 (1.394) |
  Leukocytes: Week 48: number analyzed (Participants) | 0 | 0 | 45
  Leukocytes: Week 48 |  |  | -0.25 (1.008)

31. Secondary Outcome: Change From Baseline in Hematology Parameter: Hemoglobin Values at Weeks 24 and 48
Description: Change from baseline in hematology parameter: hemoglobin values at Weeks 24 and 48 were reported.
Time Frame: as for outcome 10
Population: as for outcome 27
Measure: Mean (Standard Deviation); unit: grams per liter (g/L)
Arm/Group | INI + TAF/FTC Delayed Switch (DS1): Baseline to Week 24 | D/C/F/TAF Immediate Switch (IS1): Baseline to Week 24 | D/C/F/TAF Immediate Switch (IS): Baseline to Week 48
Number analyzed (Participants) | 43 | 42 | 45
grams per liter (g/L)
  Week 24: number analyzed (Participants) | 43 | 42 | 0
  Week 24 | -0.1 (9.98) | -1.2 (7.25) |
  Week 48: number analyzed (Participants) | 0 | 0 | 45
  Week 48 |  |  | -2.7 (7.45)

32. Secondary Outcome: Change From Baseline in Hematology Parameter: Erythrocytes Values at Weeks 24 and 48
Description: Change from baseline in hematology parameter: Erythrocytes values at Weeks 24 and 48 were reported.
Time Frame: as for outcome 10
Population: as for outcome 27
Measure: Mean (Standard Deviation); unit: 10^12 cells per liter
Arm/Group | INI + TAF/FTC Delayed Switch (DS1): Baseline to Week 24 | D/C/F/TAF Immediate Switch (IS1): Baseline to Week 24 | D/C/F/TAF Immediate Switch (IS): Baseline to Week 48
Number analyzed (Participants) | 43 | 42 | 45
10^12 cells per liter
  Week 24: number analyzed (Participants) | 43 | 42 | 0
  Week 24 | 0.05 (0.233) | -0.06 (0.257) |
  Week 48: number analyzed (Participants) | 0 | 0 | 45
  Week 48 |  |  | -0.09 (0.273)

33. Secondary Outcome: Change From Baseline in Urinalysis Parameter: Specific Gravity Values at Weeks 24 and 48
Description: Change from baseline in urinalysis parameter (specific gravity) values at Weeks 24 and 48 were reported.
Time Frame: as for outcome 10
Population: as for outcome 27
Measure: Mean (Standard Deviation); unit: kg/m^3
Arm/Group | INI + TAF/FTC Delayed Switch (DS1): Baseline to Week 24 | D/C/F/TAF Immediate Switch (IS1): Baseline to Week 24 | D/C/F/TAF Immediate Switch (IS): Baseline to Week 48
Number analyzed (Participants) | 43 | 46 | 45
kg/m^3
  Week 24: number analyzed (Participants) | 43 | 46 | 0
  Week 24 | 0.00 (0.008) | 0.00 (0.008) |
  Week 48: number analyzed (Participants) | 0 | 0 | 45
  Week 48 |  |  | 0.00 (0.009)

34. Secondary Outcome: Change From Baseline in Urinalysis Parameter: pH Values at Weeks 24 and 48
Description: Change from baseline in urinalysis parameter: pH values at Weeks 24 and 48 were reported. The pH scale measures how acidic or alkaline a substance is. The scale ranges from 0 to 14. A pH of 7 is neutral. A pH less than 7 is acidic, and a pH greater than 7 is basic. Higher the pH value, more alkaline is the substance.
Time Frame: as for outcome 10
Population: as for outcome 27
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | INI + TAF/FTC Delayed Switch (DS1): Baseline to Week 24 | D/C/F/TAF Immediate Switch (IS1): Baseline to Week 24 | D/C/F/TAF Immediate Switch (IS): Baseline to Week 48
Number analyzed (Participants) | 43 | 46 | 45
Units on a scale
  Week 24: number analyzed (Participants) | 43 | 46 | 0
  Week 24 | 0.00 (0.463) | -0.07 (0.490) |
  Week 48: number analyzed (Participants) | 0 | 0 | 45
  Week 48 |  |  | -0.06 (0.503)

35. Secondary Outcome: Number of Participants With Grade 3 and Grade 4 Laboratory Abnormalities
Description: Number of participants with grade 3 and grade 4 laboratory abnormalities were reported. Grades were assessed by Division of Acquired Immunodeficiency Syndrome (DAIDS) grading table: Grade 1: mild ; Grade 2: moderate ; Grade 3: severe ; Grade 4: potentially life-threatening ; Grade 5: death. Higher grades indicated worsening of abnormalities.
Time Frame: as for outcome 21
Population: as for outcome 21
Measure: Count of Participants; unit: Participants
Arm/Group | INI + TAF/FTC Delayed Switch (DS1): Baseline to Week 24 | D/C/F/TAF Immediate Switch (IS1): Baseline-Week 24 | D/C/F/TAF Immediate Switch (IS2): Week 25-48 | INI + TAF/FTC to D/C/F/TAF Delayed Switch (DS2): Week 25-Week 48
Number analyzed (Participants) | 50 | 53 | 49 | 46
Participants | 1 | 2 | 1 | 1

36. Secondary Outcome: Percentage of Participants With Confirmed Virologic Rebound at Weeks 24 and 48
Description: Percentage of participants with confirmed virologic rebound at Weeks 24 and 48 was reported. Virologic rebound defined as when 2 consecutive HIV-1 RNA values >=200 copies/mL at a scheduled or unscheduled visit.
Time Frame: as for outcome 19
Population: The ITT analysis set included all the participants who were randomized and received at least 1 dose of treatment subsequent to randomization in the study. Here, 'n' (number analyzed) is defined as participants analyzed at specified timepoints. Here, n=0 signifies that participants were not planned to be analyzed at those timepoints in the respective arms.
Measure: Number; unit: Percentage of Participants
Arm/Group | INI + TAF/FTC Delayed Switch (DS1): Baseline to Week 24 | D/C/F/TAF Immediate Switch (IS1): Baseline to Week 24 | D/C/F/TAF Immediate Switch (IS): Baseline to Week 48
Number analyzed (Participants) | 50 | 53 | 53
Percentage of Participants
  Week 24: number analyzed (Participants) | 50 | 53 | 0
  Week 24 | 4.0 | 0 |
  Week 48: number analyzed (Participants) | 0 | 0 | 53
  Week 48 |  |  | 0

37. Secondary Outcome: Percentage of Participants With Virologic Response (HIV-1 RNA<50 Copies/mL) at Weeks 24 and 48
Description: Percentage of participants with virologic response (HIV-1 RNA<50 copies/mL) at Weeks 24 and 48 was reported.
Time Frame: as for outcome 19
Population: as for outcome 36
Measure: Number; unit: Percentage of Participants
Arm/Group | INI + TAF/FTC Delayed Switch (DS1): Baseline to Week 24 | D/C/F/TAF Immediate Switch (IS1): Baseline to Week 24 | D/C/F/TAF Immediate Switch (IS): Baseline to Week 48
Number analyzed (Participants) | 50 | 53 | 53
Percentage of Participants
  Week 24: number analyzed (Participants) | 50 | 53 | 0
  Week 24 | 80.0 | 90.6 |
  Week 48: number analyzed (Participants) | 0 | 0 | 53
  Week 48 |  |  | 81.1

38. Secondary Outcome: Percentage of Participants With Virologic Failure (HIV-1 RNA >=50 Copies/mL) at Weeks 24 and 48
Description: Percentage of participants with virologic failure (HIV-1 RNA >=50 copies/mL) at Weeks 24 and 48 was reported.
Time Frame: as for outcome 19
Population: as for outcome 36
Measure: Number; unit: Percentage of Participants
Arm/Group | INI + TAF/FTC Delayed Switch (DS1): Baseline to Week 24 | D/C/F/TAF Immediate Switch (IS1): Baseline to Week 24 | D/C/F/TAF Immediate Switch (IS): Baseline to Week 48
Number analyzed (Participants) | 50 | 53 | 53
Percentage of Participants
  Week 24: number analyzed (Participants) | 50 | 53 | 0
  Week 24 | 10.0 | 0 |
  Week 48: number analyzed (Participants) | 0 | 0 | 53
  Week 48 |  |  | 3.8

39. Secondary Outcome: Percentage of Participants With Virologic Response (HIV-1 RNA<200 Copies/mL) at Weeks 24 and 48
Description: Percentage of participants with virologic response (HIV-1 RNA<200 copies/mL) at Week 24 and 48 was reported.
Time Frame: as for outcome 19
Population: as for outcome 36
Measure: Number; unit: Percentage of Participants
Arm/Group | INI + TAF/FTC Delayed Switch (DS1): Baseline to Week 24 | D/C/F/TAF Immediate Switch (IS1): Baseline to Week 24 | D/C/F/TAF Immediate Switch (IS): Baseline to Week 48
Number analyzed (Participants) | 50 | 53 | 53
Percentage of Participants
  Week 24: number analyzed (Participants) | 50 | 53 | 0
  Week 24 | 86.0 | 90.6 |
  Week 48: number analyzed (Participants) | 0 | 0 | 53
  Week 48 |  |  | 84.9

40. Secondary Outcome: Percentage of Participants With Virologic Failure (HIV-1 RNA >=200 Copies/mL) at Weeks 24 and 48
Description: Percentage of participants with virologic failure (HIV-1 RNA >=200 copies/mL) at Weeks 24 and 48 was reported.
Time Frame: as for outcome 19
Population: as for outcome 36
Measure: Number; unit: Percentage of Participants
Arm/Group | INI + TAF/FTC Delayed Switch (DS1): Baseline to Week 24 | D/C/F/TAF Immediate Switch (IS1): Baseline to Week 24 | D/C/F/TAF Immediate Switch (IS): Baseline to Week 48
Number analyzed (Participants) | 50 | 53 | 53
Percentage of Participants
  Week 24: number analyzed (Participants) | 50 | 53 | 0
  Week 24 | 4.0 | 0 |
  Week 48: number analyzed (Participants) | 0 | 0 | 53
  Week 48 |  |  | 0

41. Secondary Outcome: Change From Baseline in Cluster of Differentiation-4 (CD4+) Cell Count at Weeks 24 and 48
Description: Change from baseline in CD4+ cell count at Weeks 24 and 48 were reported.
Time Frame: as for outcome 10
Population: as for outcome 27
Measure: Median (Inter-Quartile Range); unit: Cells per cubic millimeter (cells/mm^3)
Arm/Group | INI + TAF/FTC Delayed Switch (DS1): Baseline to Week 24 | D/C/F/TAF Immediate Switch (IS1): Baseline to Week 24 | D/C/F/TAF Immediate Switch (IS): Baseline to Week 48
Number analyzed (Participants) | 43 | 42 | 43
Cells per cubic millimeter (cells/mm^3)
  Week 24: number analyzed (Participants) | 43 | 42 | 0
  Week 24 | 9.0 [-54.0 to 95.0] | 61.0 [34.0 to 89.0] |
  Week 48: number analyzed (Participants) | 0 | 0 | 43
  Week 48 |  |  | -41.0 [-121.0 to 127.0]

42. Secondary Outcome: Percentage of Participants Who Had Bothersome Symptoms (Scores of 1, 2, 3 or 4) Across All Items of the HIV-Symptom Index (HIV-SI) at Weeks 24 and 48
Description: Percentage of participants who had bothersome symptoms (scores of 1, 2, 3 or 4) across all items of the HIV-SI at Weeks 24 and 48 were reported. HIV-SI is a validated PRO instrument to assess 20 common HIV symptoms: fatigue/loss of energy, difficulty sleeping, nervous/anxious, diarrhea/loose bowels, changes in body composition, feeling sad/down/depressed, bloating/pain/gas in stomach, muscle aches/joint pain, problems with sex, trouble remembering, headaches, pain/numbness/tingling in hands/feet, skin problems/rash/itching, cough/trouble breathing, fever/chills/sweats, dizzy/lightheadedness, body weight loss/wasting, nausea/vomiting, hair loss/changes, and loss of appetite/food taste. Symptoms were rated using a 5-point Likert scale: 0: I don't have this symptom; 1: I have this symptom and it doesn't bother me; 2: I have this symptom and it bothers me a little; 3: I have this symptom and it bothers me; 4: I have this symptom and it bothers me a lot. Higher score refers more symptoms.
Time Frame: as for outcome 10
Population: as for outcome 7
Measure: Number; unit: Percentage of Participants
Arm/Group | INI + TAF/FTC Delayed Switch (DS1): Baseline to Week 24 | D/C/F/TAF Immediate Switch (IS1): Baseline to Week 24 | D/C/F/TAF Immediate Switch (IS): Baseline to Week 48
Number analyzed (Participants) | 49 | 44 | 46
Percentage of Participants
  Fatigue or loss of energy?: Baseline: number analyzed (Participants) | 49 | 0 | 46
  Fatigue or loss of energy?: Baseline | 61.2 |  | 43.5
  Fatigue or loss of energy?: Week 24: number analyzed (Participants) | 44 | 44 | 0
  Fatigue or loss of energy?: Week 24 | 54.5 | 47.7 |
  Fatigue or loss of energy?: Week 48: number analyzed (Participants) | 0 | 0 | 42
  Fatigue or loss of energy?: Week 48 |  |  | 42.9
  Fever, chills or sweats?: Baseline: number analyzed (Participants) | 49 | 0 | 46
  Fever, chills or sweats?: Baseline | 26.5 |  | 13.0
  Fever, chills or sweats?: Week 24: number analyzed (Participants) | 44 | 44 | 0
  Fever, chills or sweats?: Week 24 | 20.5 | 11.4 |
  Fever, chills or sweats?: Week 48: number analyzed (Participants) | 0 | 0 | 42
  Fever, chills or sweats?: Week 48 |  |  | 16.7
  Feeling dizzy or lightheaded?: Baseline: number analyzed (Participants) | 49 | 0 | 46
  Feeling dizzy or lightheaded?: Baseline | 28.6 |  | 8.7
  Feeling dizzy or lightheaded?: Week 24: number analyzed (Participants) | 44 | 44 | 0
  Feeling dizzy or lightheaded?: Week 24 | 29.5 | 13.6 |
  Feeling dizzy or lightheaded?: Week 48: number analyzed (Participants) | 0 | 0 | 42
  Feeling dizzy or lightheaded?: Week 48 |  |  | 21.4
  Pain, numbness or tingling in the hands or feet?: Baseline: number analyzed (Participants) | 49 | 0 | 46
  Pain, numbness or tingling in the hands or feet?: Baseline | 42.9 |  | 30.4
  Pain, numbness or tingling in the hands or feet?: Week 24: number analyzed (Participants) | 44 | 44 | 0
  Pain, numbness or tingling in the hands or feet?: Week 24 | 38.6 | 20.5 |
  Pain, numbness or tingling in the hands or feet?: Week 48: number analyzed (Participants) | 0 | 0 | 42
  Pain, numbness or tingling in the hands or feet?: Week 48 |  |  | 33.3
  Trouble remembering? : Baseline: number analyzed (Participants) | 49 | 0 | 46
  Trouble remembering? : Baseline | 53.1 |  | 32.6
  Trouble remembering? : Week 24: number analyzed (Participants) | 44 | 44 | 0
  Trouble remembering? : Week 24 | 38.6 | 34.1 |
  Trouble remembering? : Week 48: number analyzed (Participants) | 0 | 0 | 42
  Trouble remembering? : Week 48 |  |  | 38.1
  Nausea or vomiting?: Baseline: number analyzed (Participants) | 49 | 0 | 46
  Nausea or vomiting?: Baseline | 14.3 |  | 4.3
  Nausea or vomiting?: Week 24: number analyzed (Participants) | 40 | 44 | 0
  Nausea or vomiting?: Week 24 | 11.4 | 13.6 |
  Nausea or vomiting?: Week 48: number analyzed (Participants) | 0 | 0 | 42
  Nausea or vomiting?: Week 48 |  |  | 9.5
  Diarrhea or loose bowel movements?: Baseline: number analyzed (Participants) | 49 | 0 | 46
  Diarrhea or loose bowel movements?: Baseline | 32.7 |  | 8.7
  Diarrhea or loose bowel movements?: Week 24: number analyzed (Participants) | 44 | 44 | 0
  Diarrhea or loose bowel movements?: Week 24 | 27.3 | 31.8 |
  Diarrhea or loose bowel movements?: Week 48: number analyzed (Participants) | 0 | 0 | 42
  Diarrhea or loose bowel movements?: Week 48 |  |  | 21.4
  Felt sad, down or depressed?: Baseline: number analyzed (Participants) | 49 | 0 | 46
  Felt sad, down or depressed?: Baseline | 59.2 |  | 39.1
  Felt sad, down or depressed?: Week 24: number analyzed (Participants) | 44 | 44 | 0
  Felt sad, down or depressed?: Week 24 | 52.3 | 34.1 |
  Felt sad, down or depressed?: Week 48: number analyzed (Participants) | 0 | 0 | 42
  Felt sad, down or depressed?: Week 48 |  |  | 40.5
  Felt nervous or anxious?: Baseline: number analyzed (Participants) | 49 | 0 | 46
  Felt nervous or anxious?: Baseline | 55.1 |  | 32.6
  Felt nervous or anxious?: Week 24: number analyzed (Participants) | 44 | 44 | 0
  Felt nervous or anxious?: Week 24 | 43.2 | 38.6 |
  Felt nervous or anxious?: Week 48: number analyzed (Participants) | 0 | 0 | 42
  Felt nervous or anxious?: Week 48 |  |  | 47.6
  Difficulty falling or staying asleep? : Baseline: number analyzed (Participants) | 49 | 0 | 46
  Difficulty falling or staying asleep? : Baseline | 59.2 |  | 45.7
  Difficulty falling or staying asleep?: Week 24: number analyzed (Participants) | 44 | 44 | 0
  Difficulty falling or staying asleep?: Week 24 | 56.8 | 52.3 |
  Difficulty falling or staying asleep?: Week 48: number analyzed (Participants) | 0 | 0 | 42
  Difficulty falling or staying asleep?: Week 48 |  |  | 54.8
  Skin problems, such as rash, dryness or itching?: Baseline: number analyzed (Participants) | 49 | 0 | 46
  Skin problems, such as rash, dryness or itching?: Baseline | 34.7 |  | 34.8
  Skin problems, such as rash, dryness or itching?: Week 24: number analyzed (Participants) | 44 | 44 | 0
  Skin problems, such as rash, dryness or itching?: Week 24 | 31.8 | 22.7 |
  Skin problems, such as rash, dryness or itching?: Week 48: number analyzed (Participants) | 0 | 0 | 42
  Skin problems, such as rash, dryness or itching?: Week 48 |  |  | 38.1
  Cough or trouble catching your breath?: Baseline: number analyzed (Participants) | 49 | 0 | 46
  Cough or trouble catching your breath?: Baseline | 36.7 |  | 10.9
  Cough or trouble catching your breath?: Week 24: number analyzed (Participants) | 44 | 44 | 0
  Cough or trouble catching your breath?: Week 24 | 22.7 | 18.2 |
  Cough or trouble catching your breath?: Week 48: number analyzed (Participants) | 0 | 0 | 42
  Cough or trouble catching your breath?: Week 48 |  |  | 9.5
  Headache? : Baseline: number analyzed (Participants) | 49 | 0 | 46
  Headache? : Baseline | 36.7 |  | 19.6
  Headache? : Week 24: number analyzed (Participants) | 44 | 44 | 0
  Headache? : Week 24 | 18.2 | 22.7 |
  Headache? : Week 48: number analyzed (Participants) | 0 | 0 | 42
  Headache? : Week 48 |  |  | 26.2
  Loss of appetite or a change in the taste of food?: Baseline: number analyzed (Participants) | 49 | 0 | 46
  Loss of appetite or a change in the taste of food?: Baseline | 30.6 |  | 10.9
  Loss of appetite or a change in the taste of food?: Week 24: number analyzed (Participants) | 44 | 44 | 0
  Loss of appetite or a change in the taste of food?: Week 24 | 20.5 | 22.7 |
  Loss of appetite or a change in the taste of food?: Week 48: number analyzed (Participants) | 0 | 0 | 42
  Loss of appetite or a change in the taste of food?: Week 48 |  |  | 21.4
  Bloating, pain or gas in your stomach?: Baseline: number analyzed (Participants) | 49 | 0 | 46
  Bloating, pain or gas in your stomach?: Baseline | 40.8 |  | 39.1
  Bloating, pain or gas in your stomach?: Week 24: number analyzed (Participants) | 44 | 44 | 0
  Bloating, pain or gas in your stomach?: Week 24 | 40.9 | 38.6 |
  Bloating, pain or gas in your stomach?: Week 48: number analyzed (Participants) | 0 | 0 | 42
  Bloating, pain or gas in your stomach?: Week 48 |  |  | 33.3
  Muscle aches or joint pain?: Baseline: number analyzed (Participants) | 49 | 0 | 46
  Muscle aches or joint pain?: Baseline | 53.1 |  | 34.8
  Muscle aches or joint pain?: Week 24: number analyzed (Participants) | 44 | 44 | 0
  Muscle aches or joint pain?: Week 24 | 45.5 | 38.6 |
  Muscle aches or joint pain?: Week 48: number analyzed (Participants) | 0 | 0 | 42
  Muscle aches or joint pain?: Week 48 |  |  | 42.9
  Problems with having sex, such as loss of interest or lack of satisfaction?: Baseline: number analyzed (Participants) | 49 | 0 | 46
  Problems with having sex, such as loss of interest or lack of satisfaction?: Baseline | 42.9 |  | 39.1
  Problems with having sex, such as loss of interest or lack of satisfaction?: Week 24: number analyzed (Participants) | 44 | 44 | 0
  Problems with having sex, such as loss of interest or lack of satisfaction?: Week 24 | 22.7 | 38.6 |
  Problems with having sex, such as loss of interest or lack of satisfaction?: Week 48: number analyzed (Participants) | 0 | 0 | 42
  Problems with having sex, such as loss of interest or lack of satisfaction?: Week 48 |  |  | 26.2
  Changes in the way your body looks such as fat deposits or weight gain?: Baseline: number analyzed (Participants) | 49 | 0 | 46
  Changes in the way your body looks such as fat deposits or weight gain?: Baseline | 71.4 |  | 71.7
  Changes in the way your body looks such as fat deposits or weight gain?: Week 24: number analyzed (Participants) | 44 | 44 | 0
  Changes in the way your body looks such as fat deposits or weight gain?: Week 24 | 70.5 | 63.6 |
  Changes in the way your body looks such as fat deposits or weight gain?: Week 48: number analyzed (Participants) | 0 | 0 | 42
  Changes in the way your body looks such as fat deposits or weight gain?: Week 48 |  |  | 59.5
  Problems with weight loss or wasting?: Baseline: number analyzed (Participants) | 49 | 0 | 46
  Problems with weight loss or wasting?: Baseline | 32.7 |  | 17.4
  Problems with weight loss or wasting?: Week 24: number analyzed (Participants) | 44 | 44 | 0
  Problems with weight loss or wasting?: Week 24 | 29.5 | 15.9 |
  Problems with weight loss or wasting?: Week 48: number analyzed (Participants) | 0 | 0 | 42
  Problems with weight loss or wasting?: Week 48 |  |  | 26.2
  Hair loss or changes in the way your hair looks?: Baseline: number analyzed (Participants) | 49 | 0 | 46
  Hair loss or changes in the way your hair looks?: Baseline | 26.5 |  | 19.6
  Hair loss or changes in the way your hair looks?: Week 24: number analyzed (Participants) | 44 | 44 | 0
  Hair loss or changes in the way your hair looks?: Week 24 | 20.5 | 34.1 |
  Hair loss or changes in the way your hair looks?: Week 48: number analyzed (Participants) | 0 | 0 | 42
  Hair loss or changes in the way your hair looks?: Week 48 |  |  | 23.8

43. Secondary Outcome: Percentage of Participants Who Had Any Symptoms (Scores of 1, 2, 3 or 4) Across All Items of the HIV-Symptom Index (HIV-SI) at Weeks 24 and 48
Description: Percentage of participants who had any symptoms (scores of 1, 2, 3 or 4) across all items of the HIV-SI at Weeks 24 and 48 were reported. HIV-SI is a validated PRO instrument to assess 20 common HIV symptoms: fatigue/loss of energy, difficulty sleeping, nervous/anxious, diarrhea/loose bowels, changes in body composition, feeling sad/down/depressed, bloating/pain/gas in stomach, muscle aches/joint pain, problems with sex, trouble remembering, headaches, pain/numbness/tingling in hands/feet, skin problems/rash/itching, cough/trouble breathing, fever/chills/sweats, dizzy/lightheadedness, body weight loss/wasting, nausea/vomiting, hair loss/changes, and loss of appetite/food taste. Symptoms were rated using a 5-point Likert scale: 0: I don't have this symptom; 1: I have this symptom and it doesn't bother me; 2: I have this symptom and it bothers me a little; 3: I have this symptom and it bothers me; 4: I have this symptom and it bothers me a lot. Higher score refers more symptoms.
Time Frame: as for outcome 10
Population: as for outcome 7
Measure: Number; unit: Percentage of Participants
Arm/Group | INI + TAF/FTC Delayed Switch (DS1): Baseline to Week 24 | D/C/F/TAF Immediate Switch (IS1): Baseline to Week 24 | D/C/F/TAF Immediate Switch (IS): Baseline to Week 48
Number analyzed (Participants) | 49 | 44 | 46
Percentage of Participants
  Fatigue or loss of energy?: Baseline: number analyzed (Participants) | 49 | 0 | 46
  Fatigue or loss of energy?: Baseline | 73.5 |  | 45.7
  Fatigue or loss of energy?: Week 24: number analyzed (Participants) | 44 | 44 | 0
  Fatigue or loss of energy?: Week 24 | 61.4 | 59.1 |
  Fatigue or loss of energy?: Week 48: number analyzed (Participants) | 0 | 0 | 42
  Fatigue or loss of energy?: Week 48 |  |  | 47.6
  Fever, chills or sweats?: Baseline: number analyzed (Participants) | 49 | 0 | 46
  Fever, chills or sweats?: Baseline | 34.7 |  | 17.4
  Fever, chills or sweats?: Week 24: number analyzed (Participants) | 44 | 44 | 0
  Fever, chills or sweats?: Week 24 | 29.5 | 20.5 |
  Fever, chills or sweats?: Week 48: number analyzed (Participants) | 0 | 0 | 42
  Fever, chills or sweats?: Week 48 |  |  | 26.2
  Feeling dizzy or lightheaded?: Baseline: number analyzed (Participants) | 49 | 0 | 46
  Feeling dizzy or lightheaded?: Baseline | 34.7 |  | 17.4
  Feeling dizzy or lightheaded?: Week 24: number analyzed (Participants) | 44 | 44 | 0
  Feeling dizzy or lightheaded?: Week 24 | 36.4 | 27.3 |
  Feeling dizzy or lightheaded?: Week 48: number analyzed (Participants) | 0 | 0 | 42
  Feeling dizzy or lightheaded?: Week 48 |  |  | 28.6
  Pain, numbness or tingling in the hands or feet?: Baseline: number analyzed (Participants) | 49 | 0 | 46
  Pain, numbness or tingling in the hands or feet?: Baseline | 53.1 |  | 43.5
  Pain, numbness or tingling in the hands or feet?: Week 24: number analyzed (Participants) | 44 | 44 | 0
  Pain, numbness or tingling in the hands or feet?: Week 24 | 47.7 | 34.1 |
  Pain, numbness or tingling in the hands or feet?: Week 48: number analyzed (Participants) | 0 | 0 | 42
  Pain, numbness or tingling in the hands or feet?: Week 48 |  |  | 42.9
  Trouble remembering? : Baseline: number analyzed (Participants) | 49 | 0 | 46
  Trouble remembering? : Baseline | 59.2 |  | 47.8
  Trouble remembering? : Week 24: number analyzed (Participants) | 44 | 44 | 0
  Trouble remembering? : Week 24 | 47.7 | 45.5 |
  Trouble remembering? : Week 48: number analyzed (Participants) | 0 | 0 | 42
  Trouble remembering? : Week 48 |  |  | 47.6
  Nausea or vomiting?: Baseline: number analyzed (Participants) | 49 | 0 | 46
  Nausea or vomiting?: Baseline | 24.5 |  | 8.7
  Nausea or vomiting?: Week 24: number analyzed (Participants) | 40 | 44 | 0
  Nausea or vomiting?: Week 24 | 15.9 | 18.2 |
  Nausea or vomiting?: Week 48: number analyzed (Participants) | 0 | 0 | 42
  Nausea or vomiting?: Week 48 |  |  | 16.7
  Diarrhea or loose bowel movements?: Baseline: number analyzed (Participants) | 49 | 0 | 46
  Diarrhea or loose bowel movements?: Baseline | 46.9 |  | 17.4
  Diarrhea or loose bowel movements?: Week 24: number analyzed (Participants) | 44 | 44 | 0
  Diarrhea or loose bowel movements?: Week 24 | 36.4 | 43.2 |
  Diarrhea or loose bowel movements?: Week 48: number analyzed (Participants) | 0 | 0 | 42
  Diarrhea or loose bowel movements?: Week 48 |  |  | 35.7
  Felt sad, down or depressed?: Baseline: number analyzed (Participants) | 49 | 0 | 46
  Felt sad, down or depressed?: Baseline | 73.5 |  | 54.3
  Felt sad, down or depressed?: Week 24: number analyzed (Participants) | 44 | 44 | 0
  Felt sad, down or depressed?: Week 24 | 61.4 | 50.0 |
  Felt sad, down or depressed?: Week 48: number analyzed (Participants) | 0 | 0 | 42
  Felt sad, down or depressed?: Week 48 |  |  | 47.6
  Felt nervous or anxious?: Baseline: number analyzed (Participants) | 49 | 0 | 46
  Felt nervous or anxious?: Baseline | 63.3 |  | 63.0
  Felt nervous or anxious?: Week 24: number analyzed (Participants) | 44 | 44 | 0
  Felt nervous or anxious?: Week 24 | 59.1 | 50.0 |
  Felt nervous or anxious?: Week 48: number analyzed (Participants) | 0 | 0 | 42
  Felt nervous or anxious?: Week 48 |  |  | 54.8
  Difficulty falling or staying asleep? : Baseline: number analyzed (Participants) | 49 | 0 | 46
  Difficulty falling or staying asleep? : Baseline | 65.3 |  | 50.0
  Difficulty falling or staying asleep?: Week 24: number analyzed (Participants) | 44 | 44 | 0
  Difficulty falling or staying asleep?: Week 24 | 63.6 | 61.4 |
  Difficulty falling or staying asleep?: Week 48: number analyzed (Participants) | 0 | 0 | 42
  Difficulty falling or staying asleep?: Week 48 |  |  | 64.3
  Skin problems, such as rash, dryness or itching?: Baseline: number analyzed (Participants) | 49 | 0 | 46
  Skin problems, such as rash, dryness or itching?: Baseline | 42.9 |  | 41.3
  Skin problems, such as rash, dryness or itching?: Week 24: number analyzed (Participants) | 44 | 44 | 0
  Skin problems, such as rash, dryness or itching?: Week 24 | 40.9 | 34.1 |
  Skin problems, such as rash, dryness or itching?: Week 48: number analyzed (Participants) | 0 | 0 | 42
  Skin problems, such as rash, dryness or itching?: Week 48 |  |  | 45.2
  Cough or trouble catching your breath?: Baseline: number analyzed (Participants) | 49 | 0 | 46
  Cough or trouble catching your breath?: Baseline | 46.9 |  | 19.6
  Cough or trouble catching your breath?: Week 24: number analyzed (Participants) | 44 | 44 | 0
  Cough or trouble catching your breath?: Week 24 | 29.5 | 31.8 |
  Cough or trouble catching your breath?: Week 48: number analyzed (Participants) | 0 | 0 | 42
  Cough or trouble catching your breath?: Week 48 |  |  | 21.4
  Headache? : Baseline: number analyzed (Participants) | 49 | 0 | 46
  Headache? : Baseline | 46.9 |  | 30.4
  Headache? : Week 24: number analyzed (Participants) | 44 | 44 | 0
  Headache? : Week 24 | 29.5 | 29.5 |
  Headache? : Week 48: number analyzed (Participants) | 0 | 0 | 42
  Headache? : Week 48 |  |  | 38.1
  Loss of appetite or a change in the taste of food?: Baseline: number analyzed (Participants) | 49 | 0 | 46
  Loss of appetite or a change in the taste of food?: Baseline | 36.7 |  | 21.7
  Loss of appetite or a change in the taste of food?: Week 24: number analyzed (Participants) | 44 | 44 | 0
  Loss of appetite or a change in the taste of food?: Week 24 | 29.5 | 25.0 |
  Loss of appetite or a change in the taste of food?: Week 48: number analyzed (Participants) | 0 | 0 | 42
  Loss of appetite or a change in the taste of food?: Week 48 |  |  | 31.0
  Bloating, pain or gas in your stomach?: Baseline: number analyzed (Participants) | 49 | 0 | 46
  Bloating, pain or gas in your stomach?: Baseline | 46.9 |  | 56.5
  Bloating, pain or gas in your stomach?: Week 24: number analyzed (Participants) | 44 | 44 | 0
  Bloating, pain or gas in your stomach?: Week 24 | 45.5 | 54.5 |
  Bloating, pain or gas in your stomach?: Week 48: number analyzed (Participants) | 0 | 0 | 42
  Bloating, pain or gas in your stomach?: Week 48 |  |  | 52.4
  Muscle aches or joint pain?: Baseline: number analyzed (Participants) | 49 | 0 | 46
  Muscle aches or joint pain?: Baseline | 57.1 |  | 43.5
  Muscle aches or joint pain?: Week 24: number analyzed (Participants) | 44 | 44 | 0
  Muscle aches or joint pain?: Week 24 | 47.7 | 43.2 |
  Muscle aches or joint pain?: Week 48: number analyzed (Participants) | 0 | 0 | 42
  Muscle aches or joint pain?: Week 48 |  |  | 52.4
  Problems with having sex, such as loss of interest or lack of satisfaction?: Baseline: number analyzed (Participants) | 49 | 0 | 46
  Problems with having sex, such as loss of interest or lack of satisfaction?: Baseline | 51.0 |  | 47.8
  Problems with having sex, such as loss of interest or lack of satisfaction?: Week 24: number analyzed (Participants) | 44 | 44 | 0
  Problems with having sex, such as loss of interest or lack of satisfaction?: Week 24 | 31.8 | 52.3 |
  Problems with having sex, such as loss of interest or lack of satisfaction?: Week 48: number analyzed (Participants) | 0 | 0 | 42
  Problems with having sex, such as loss of interest or lack of satisfaction?: Week 48 |  |  | 40.5
  Changes in the way your body looks such as fat deposits or weight gain?: Baseline: number analyzed (Participants) | 49 | 0 | 46
  Changes in the way your body looks such as fat deposits or weight gain?: Baseline | 77.6 |  | 80.4
  Changes in the way your body looks such as fat deposits or weight gain?: Week 24: number analyzed (Participants) | 44 | 44 | 0
  Changes in the way your body looks such as fat deposits or weight gain?: Week 24 | 77.3 | 72.7 |
  Changes in the way your body looks such as fat deposits or weight gain?: Week 48: number analyzed (Participants) | 0 | 0 | 42
  Changes in the way your body looks such as fat deposits or weight gain?: Week 48 |  |  | 76.2
  Problems with weight loss or wasting?: Baseline: number analyzed (Participants) | 49 | 0 | 46
  Problems with weight loss or wasting?: Baseline | 36.7 |  | 21.7
  Problems with weight loss or wasting?: Week 24: number analyzed (Participants) | 44 | 44 | 0
  Problems with weight loss or wasting?: Week 24 | 38.6 | 25.0 |
  Problems with weight loss or wasting?: Week 48: number analyzed (Participants) | 0 | 0 | 42
  Problems with weight loss or wasting?: Week 48 |  |  | 35.7
  Hair loss or changes in the way your hair looks?: Baseline: number analyzed (Participants) | 49 | 0 | 46
  Hair loss or changes in the way your hair looks?: Baseline | 34.7 |  | 26.1
  Hair loss or changes in the way your hair looks?: Week 24: number analyzed (Participants) | 44 | 44 | 0
  Hair loss or changes in the way your hair looks?: Week 24 | 27.3 | 38.6 |
  Hair loss or changes in the way your hair looks?: Week 48: number analyzed (Participants) | 0 | 0 | 42
  Hair loss or changes in the way your hair looks?: Week 48 |  |  | 35.7

44. Secondary Outcome: Number of Participants With Each Bothersome Symptom of the HIV-SI Adjusting for Baseline Variables at Weeks 24 and 48
Description: Number of participants With each bothersome symptom of the HIV-SI adjusting for baseline variables at Weeks 24 and 48 were reported.
Time Frame: as for outcome 19
Population: The ITT analysis set included all the participants who were randomized and received at least 1 dose of treatment subsequent to randomization in the study. Here, n=0 signifies that participants were not planned to be analyzed at those timepoints in the respective arms. Here, n=0 signifies that participants were not planned to be analyzed at those timepoints in the respective arms.
Measure: Count of Participants; unit: Participants
Arm/Group | INI + TAF/FTC Delayed Switch (DS1): Baseline to Week 24 | D/C/F/TAF Immediate Switch (IS1): Baseline to Week 24 | D/C/F/TAF Immediate Switch (IS): Baseline to Week 48
Number analyzed (Participants) | 50 | 53 | 53
Participants
  Week 24: number analyzed (Participants) | 50 | 53 | 0
  Week 24 | 44 | 44 |
  Week 48: number analyzed (Participants) | 0 | 0 | 53
  Week 48 |  |  | 42

45. Secondary Outcome: Percentage of Participants With Patient Global Impression of Change (PGIC) Scale Score at Weeks 24 and 48
Description: Percentage of participants with PGIC scale score at Weeks 24 and 48 were reported. The PGI-C was a patient reported outcome (PRO) where participants rated using a 7-point scale ranging from 1 to 7 where 1 indicates "very much improved", 2 indicates "much improved', 3 indicates "minimally improved", 4 indicates "No change", 5 indicates "minimally worse", 6 indicates "Much worse" and 7 indicates "Very much worse".
Time Frame: as for outcome 19
Population: as for outcome 6
Measure: Number; unit: Percentage of Participants
Arm/Group | INI + TAF/FTC Delayed Switch (DS1): Baseline to Week 24 | D/C/F/TAF Immediate Switch (IS1): Baseline to Week 24 | D/C/F/TAF Immediate Switch (IS): Baseline to Week 48
Number analyzed (Participants) | 44 | 41 | 42
Percentage of Participants
  Very Much Improved: Week 24: number analyzed (Participants) | 44 | 41 | 0
  Very Much Improved: Week 24 | 11.4 | 4.9 |
  Much Improved: Week 24: number analyzed (Participants) | 44 | 41 | 0
  Much Improved: Week 24 | 13.6 | 22.0 |
  Minimally Improved: Week 24: number analyzed (Participants) | 44 | 41 | 0
  Minimally Improved: Week 24 | 18.2 | 19.5 |
  No Change: Week 24: number analyzed (Participants) | 44 | 41 | 0
  No Change: Week 24 | 52.3 | 19.5 |
  Minimally Worse: Week 24: number analyzed (Participants) | 44 | 41 | 0
  Minimally Worse: Week 24 | 0 | 7.3 |
  Much Worse: Week 24: number analyzed (Participants) | 44 | 41 | 0
  Much Worse: Week 24 | 2.3 | 4.9 |
  Very Much Worse: Week 24: number analyzed (Participants) | 44 | 41 | 0
  Very Much Worse: Week 24 | 2.3 | 0 |
  Very Much Improved: Week 48: number analyzed (Participants) | 0 | 0 | 42
  Very Much Improved: Week 48 |  |  | 11.9
  Much Improved: Week 48: number analyzed (Participants) | 0 | 0 | 42
  Much Improved: Week 48 |  |  | 16.7
  Minimally Improved: Week 48: number analyzed (Participants) | 0 | 0 | 42
  Minimally Improved: Week 48 |  |  | 26.2
  No Change: Week 48: number analyzed (Participants) | 0 | 0 | 42
  No Change: Week 48 |  |  | 31.0
  Minimally Worse: Week 48: number analyzed (Participants) | 0 | 0 | 42
  Minimally Worse: Week 48 |  |  | 9.5
  Much Worse: Week 48: number analyzed (Participants) | 0 | 0 | 42
  Much Worse: Week 48 |  |  | 2.4
  Very Much Worse: Week 48: number analyzed (Participants) | 0 | 0 | 42
  Very Much Worse: Week 48 |  |  | 2.4

46. Secondary Outcome: Adherence Rate to Treatment at Weeks 4, 12, 24, 36, and 48
Description: Adherence rate to treatment at Weeks 4, 12, 24, 36 and 48 were reported. Adherence rates were reported according to the percentage of participants missing 0, 1, 2, 3 or 4 doses as 100%, 75%, 50%, 25%, and 0%, respectively, using participant self-report 4-day recall at Weeks 4, 12, 24, 36, and 48.
Time Frame: Weeks 4, 12, 24, 36 and 48
Population: as for outcome 6
Measure: Number; unit: Percentage of Participants
Arm/Group | INI + TAF/FTC Delayed Switch (DS1): Baseline to Week 24 | D/C/F/TAF Immediate Switch (IS1): Baseline to Week 24 | D/C/F/TAF Immediate Switch (IS): Baseline to Week 48
Number analyzed (Participants) | 43 | 53 | 47
Percentage of Participants
  100%: Week 4: number analyzed (Participants) | 42 | 53 | 0
  100%: Week 4 | 92.9 | 90.6 |
  75%: Week 4: number analyzed (Participants) | 42 | 53 | 0
  75%: Week 4 | 7.1 | 9.4 |
  50%: Week 4: number analyzed (Participants) | 42 | 53 | 0
  50%: Week 4 | 0 | 0 |
  25%: Week 4: number analyzed (Participants) | 42 | 53 | 0
  25%: Week 4 | 0 | 0 |
  0%: Week 4: number analyzed (Participants) | 42 | 53 | 0
  0%: Week 4 | 0 | 0 |
  100%: Week 12: number analyzed (Participants) | 43 | 52 | 0
  100%: Week 12 | 93.0 | 90.4 |
  75%: Week 12: number analyzed (Participants) | 43 | 52 | 0
  75%: Week 12 | 4.7 | 7.7 |
  50%: Week 12: number analyzed (Participants) | 43 | 52 | 0
  50%: Week 12 | 0.0 | 0.0 |
  25%: Week 12: number analyzed (Participants) | 43 | 5 | 0
  25%: Week 12 | 2.3 | 1.9 |
  0%: Week 12: number analyzed (Participants) | 43 | 52 | 0
  0%: Week 12 | 0.0 | 0.0 |
  100%: Week 24: number analyzed (Participants) | 42 | 49 | 0
  100%: Week 24 | 95.2 | 98.0 |
  75%: Week 24: number analyzed (Participants) | 42 | 49 | 0
  75%: Week 24 | 2.4 | 4.1 |
  50%: Week 24: number analyzed (Participants) | 42 | 49 | 0
  50%: Week 24 | 2.4 | 0.0 |
  25%: Week 24: number analyzed (Participants) | 42 | 49 | 0
  25%: Week 24 | 0 | 0.0 |
  0%: Week 24: number analyzed (Participants) | 42 | 49 | 0
  0%: Week 24 | 0 | 0.0 |
  100%: Week 36: number analyzed (Participants) | 0 | 0 | 47
  100%: Week 36 |  |  | 93.6
  75%: Week 36: number analyzed (Participants) | 0 | 0 | 47
  75%: Week 36 |  |  | 6.4
  50%: Week 36: number analyzed (Participants) | 0 | 0 | 47
  50%: Week 36 |  |  | 0
  25%: Week 36: number analyzed (Participants) | 0 | 0 | 47
  25%: Week 36 |  |  | 0
  0%: Week 36: number analyzed (Participants) | 0 | 0 | 47
  0%: Week 36 |  |  | 0
  100%: Week 48: number analyzed (Participants) | 0 | 0 | 46
  100%: Week 48 |  |  | 93.5
  75%: Week 48: number analyzed (Participants) | 0 | 0 | 46
  75%: Week 48 |  |  | 2.2
  50%: Week 48: number analyzed (Participants) | 0 | 0 | 46
  50%: Week 48 |  |  | 0
  25%: Week 48: number analyzed (Participants) | 0 | 0 | 46
  25%: Week 48 |  |  | 2.2
  0%: Week 48: number analyzed (Participants) | 0 | 0 | 46
  0%: Week 48 |  |  | 2.2

ADVERSE EVENTS:
Time Frame: D/C/F/TAF Immediate Switch (IS1) and INI + TAF/FTC Delayed Switch (DS1): Baseline up to Week 24; D/C/F/TAF Immediate Switch (IS2) and INI + TAF/FTC to D/C/F/TAF Delayed Switch (DS2): Week 25 up to Week 48
Description: The safety analysis set included all randomized participants who received at least 1 dose of study intervention (that is, ITT analysis set).
Arm/Group | D/C/F/TAF Immediate Switch (IS1): Baseline-Week 24 | D/C/F/TAF Immediate Switch (IS2): Week 25-48 | INI + TAF/FTC Delayed Switch (DS1): Baseline to Week 24 | INI + TAF/FTC to D/C/F/TAF Delayed Switch (DS2): Week 25-Week 48
All-Cause Mortality (participants affected / at risk) | 0/53 | 0/49 | 1/50 | 0/46
Serious Adverse Events (participants affected / at risk) | 3/53 | 2/49 | 4/50 | 4/46
Other Adverse Events (participants affected / at risk) | 10/53 | 7/49 | 13/50 | 12/46
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | D/C/F/TAF Immediate Switch (IS1): Baseline-Week 24 (N=53) | D/C/F/TAF Immediate Switch (IS2): Week 25-48 (N=49) | INI + TAF/FTC Delayed Switch (DS1): Baseline to Week 24 (N=50) | INI + TAF/FTC to D/C/F/TAF Delayed Switch (DS2): Week 25-Week 48 (N=46)
Atrial Fibrillation (Cardiac disorders) | 0 | 0 | 0 | 1
Abdominal Pain (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Hypertransaminasaemia (Hepatobiliary disorders) | 1 | 0 | 0 | 0
COVID-19 (Infections and infestations) | 0 | 0 | 0 | 1
Orchitis (Infections and infestations) | 1 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 1 | 0 | 0
Pneumonia Viral (Infections and infestations) | 0 | 0 | 0 | 1
Overdose (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Upper Limb Fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Lumbar Spinal Stenosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Generalised Tonic-Clonic Seizure (Nervous system disorders) | 0 | 1 | 0 | 0
Drug Abuse (Psychiatric disorders) | 0 | 0 | 1 | 0
Abnormal Uterine Bleeding (Reproductive system and breast disorders) | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | D/C/F/TAF Immediate Switch (IS1): Baseline-Week 24 (N=53) | D/C/F/TAF Immediate Switch (IS2): Week 25-48 (N=49) | INI + TAF/FTC Delayed Switch (DS1): Baseline to Week 24 (N=50) | INI + TAF/FTC to D/C/F/TAF Delayed Switch (DS2): Week 25-Week 48 (N=46)
Diarrhoea (Gastrointestinal disorders) | 3 | 0 | 1 | 5
Nausea (Gastrointestinal disorders) | 3 | 0 | 1 | 3
Oedema Peripheral (General disorders) | 0 | 0 | 2 | 3
COVID-19 (Infections and infestations) | 6 | 3 | 2 | 1
Proctitis Gonococcal (Infections and infestations) | 0 | 3 | 1 | 1
Proteinuria (Renal and urinary disorders) | 0 | 1 | 3 | 2
Hypertension (Vascular disorders) | 1 | 1 | 6 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If an investigator wishes to publish information from the study, a copy of the manuscript must be provided to the sponsor for review at least 60 days before submission for publication or presentation. If requested by the sponsor in writing, the investigator will withhold such publication for up to an additional 60 days to allow for filing of a patent application.

DOCUMENTS (2):
  • Study Protocol (2022-04-29): https://cdn.clinicaltrials.gov/large-docs/37/NCT04442737/Prot_000.pdf
  • Statistical Analysis Plan (2023-03-24): https://cdn.clinicaltrials.gov/large-docs/37/NCT04442737/SAP_001.pdf